Document status: SAP Version 1.0



### STATISTICAL ANALYSIS PLAN

An open label phase 1b study to characterise the pharmacokinetic/pharmacodynamic relationship and safety of MMV367 in healthy adult participants experimentally infected with blood stage *Plasmodium falciparum* 

Protocol No.: MMV\_MMV367\_22\_01

**Product Code: MMV367** 

**PREPARED FOR:** Medicines for Malaria Venture (MMV)

ICC-Block G 3rd Floor 20, Route de Pré-Bois 1215 Geneva 15

Switzerland

Phone: +41 22 555 03 00

**PREPARED BY:** Southern Star Research

Level 1, 1 Merriwa St Gordon, NSW, 2072

Australia

**DATE OF ISSUE:** 15 June 2023

VERSION/STATUS: Version 1.0

**AUTHOR:** Locadiah Kuwanda

BM S01-A, v3.0

Statistical Analysis Plan

Effective: 17/SEP/2020 

## **SAP APPROVAL**

By my signature, I confirm that this SAP has been reviewed and has been approved for use on the MMV\_MMV367\_22\_01 study:

| Name | Title / Company | Signature | Date |
|------------------|---------------------|-----------|------|
| | Clinical Scientist | | |
| Etienne Guirou | Medicines for | | |
| | Malaria Venture | | |
| | Senior Statistician | | |
| Locadiah Kuwanda | Southern Star | | |
| | Research Pty Ltd. | | |

# Table of contents

| 1. | A | BBREVIATIONS | |
|----|--------------|----------------------------------------------|----|
| 2. | I٨ | NTRODUCTION | |
| 3. | PI | ROJECT OVERVIEW | 8 |
| | 3.1 | Study Design | 8 |
| | 3.2 | Schema | 9 |
| | 3.3 | Schedule of Activities | 10 |
| | 3.4 | Objectives | 13 |
| | 3.5 | Endpoints | 13 |
| | 3.6 | Sample Size | 14 |
| | 3.7 | Treatment Assignment and Randomisation | 14 |
| 4. | ST | TATISTICAL CONSIDERATIONS | 15 |
| | 4.1 | Data Capture | 15 |
| | 4.2 | Statistical Programming | 16 |
| 5. | A | NALYSIS SETS | 17 |
| | 5.1 | Analysis Set Descriptions | 17 |
| 6. | PI | ROTOCOL DEVIATIONS | 18 |
| 7. | Po | articipant DISPOSITION | 19 |
| | 7.1 [ | Disposition | 19 |
| | 7.2 <i>F</i> | Analysis of Population Assignment | 19 |
| 8. | D | EMOGRAPHIC AND BASELINE INFORMATION | 19 |
| | 8.1 | Demographics | 19 |
| | 8.2 | Medical History | 19 |
| | 8.3 | Prior Medications | 20 |
| | 8.4 | Drug Screen | 20 |
| | 8.5 | Alcohol Screen | 20 |
| | 8.6 | SARS-CoV-2 Screening | 20 |
| | 8.7 | Follicle Stimulating Hormone (FSH) | 20 |
| | 8.8 | Beck Depression Inventory | 20 |
| 9. | Tŀ | REATMENT EXPOSURE | 21 |
| 10 | | PRIMARY ENDPOINT ANALYSIS (PK/PD Analysis) | 21 |
| | 10.1 | Overview of methodology for PK/ PD Modelling | 21 |
| | 10.2 | Sources of Data | 21 |
| | 10.3 | Data Assembly | 21 |

| 1 | 0.4. | Methods | 22 |
|---|---|---|---|
| 1 | .0.5. | PK/PD Endpoints | 25 |
| 1 | .0.6. | Presentation of Results | 26 |
| 11. | SE | ECONDARY ENDPOINTS ANALYSIS | 26 |
| 1 | 1.1 | PD Analysis | 26 |
| 1 | 1.1.2 | Parasite clearance kinetics | 26 |
| 1 | 1.2 | PK Analysis | 30 |
| 1 | 1.3 | Safety | 32 |
| 12. | Ех | κploratory Parameters | 41 |
| 13. | CF | HANGES TO THE PLANNED ANALYSIS | 41 |
| 14. | IN | ITERIM AND FINAL ANALYSIS | 41 |
| 15. | SC | OFTWARE | 41 |
| 16. | RE | EFERENCES | 42 |
| 17. | | PPENDIX | |
| | | A. PD and PK Planned Tables, Listings and Figures | |
| | | 3. Baseline Characteristics and Safety Analysis Tables and Listings | |


#### 1. ABBREVIATIONS

ADaM Analysis Data Model Adverse Event ΑE

Adverse Event of Special Interest **AESI** 

ALP Alkaline phosphatase Alanine Aminotransferase ALT

APR28 Adequate Parasitological Response Rate at Day 28

Activated partial thromboplastin time **APTT** 

**AST** Aspartate Aminotransferase **ATC** Anatomical Therapeutic Chemical

Area Under the plasma Concentration Time Curve **AUC** 

Area under the curve from time 0 to last measurable concentration **AUC**<sub>last</sub>

**AUC**<sub>inf</sub> Area under the curve from time 0 to infinity

β-HCG β-Human Chorionic Gonadotropin **Beck Depression Inventory** BDI Bayesian Information Criteria BIC Below the Limit of Quantification BI Q

**Body Mass Index** BMI

Clinical Data Interchange Standards Consortium CDISC

Confidence Interval CI Creatine Kinase CK

CL/F **Apparent Oral Clearance** 

Maximum plasma concentration observed  $C_{max}$ 

COVID-19 Corona virus disease 2019 Clinical Research Associate CRA

CRF Case Report Form **CSR** Clinical Study Report

Common Terminology Criteria for Adverse Events CTCAE

CV% Coefficient of Variation **DBP** Diastolic Blood Pressure **Data Transfer Specification** DTS

Concentration at 50% of Maximum Effect EC50

**ECG** Electrocardiography

Electronic Case Report Form eCRF Electronic Data capture EDC

Maximum Effect **EMAX** FOS End of Study FAS Full Analysis Set

Follicle-Stimulating Hormone **FSH** 

Glucose-6-phosphate dehydrogenase G6PD

Gamma Glutamyl Transferase GGT Hepatitis B Surface Antigen **HBsAg HEENT** Head, Eyes, Ears, Nose, Throat HIV Human Immunodeficiency Virus

**Heart Rate** HR

Induced Blood Stage Malaria **IBSM** IIV Inter Individual Variability

Investigational Medicinal Product **IMP INR** International Normalized Ratio Lactate Dehydrogenase LDH Lower Limit of Quantification LLOQ

Limit of Quantification LOQ

Medical Dictionary for Regulatory Activities MedDRA


Minimum Inhibitory Concentration MIC MMV Medicines for Malaria Venture MPC90 Minimal Parasiticidal Concentration NCA Non-Compartmental Analysis

NΠ Non Detect

NLME Nonlinear Mixed Effects

BM S01-A, v3.0

Statistical Analysis Plan


PC Pharmacokinetics Concentration

PD Pharmacodynamics

Pf iRBC P.falciparum Infected Red Blood Cell pfMGET Male gametocyte-specific transcript

pfSBP-1 Ring-stage transcript

pfs25 Female gametocyte-specific transcript

PK Pharmacokinetics

PKPD Pharmacokinetic-pharmacodynamic

PN Preferred Name

PRR<sub>48</sub> Parasite Reduction Ratio Over 48 hours

PT Preferred Term

PCt<sub>1/2</sub> Parasite Clearance Half-Life

QIMRB QIMR Berghofer Medical Research Institute qPCR Quantitative Polymerase Chain Reaction

qRT-PCR Quantitative Reverse Transcriptase Polymerase Chain Reaction

QTcB Corrected QT interval with Bazett's Formula
QTcF Corrected QT interval with Fridericia's Formula

RAT Rapid Antigen Test SAE Serious Adverse Event

SAEM Stochastic Approximation Expectation Maximization

SAP Statistical Analysis Plan
SAS Statistical Analysis System
SBP Systolic Blood Pressure
SBQ Swiss BioQuant Central
SD Standard Deviation
SDRT Safety Data Review Team
SDTM Study Data Tabulation Model

SE Standard Error
SOC System Organ Class

SOP Standard Operating Procedure
SRC Safety Review Committee
SSR Southern Star Research
t<sub>1/2</sub> Elimination Half-Life

TEAE Treatment Emergent Adverse Event

T<sub>max</sub> Time to Reach Maximum Plasma Concentration

VIS Volunteer Infection Study

Vss/F Apparent Volume of Distribution at the Steady State After Single Dose

VPC Visual Predictive Check

Vz/F Apparent Volume of Distribution after Single Dose

WOCBP Women of Child Bearing Potential

WHODrug World Health Organization Drug Dictionary

 $\lambda_z$  Lambda-z: Slope of the apparent elimination phase


#### 2. INTRODUCTION

The following Statistical Analysis Plan (SAP) provides the outline for the statistical analysis of the data from the MMV\_MMV367\_22\_01 study. The SAP details the methods for statistical analysis of outcomes relating to safety, pharmacokinetics (PK), pharmacodynamics (PD), and population modelling of pharmacokinetic / pharmacodynamic (PK/PD) data arising from this clinical trial. This SAP has been developed and finalised prior to database lock and final analysis.

Planned analyses identified in this SAP may be included in the clinical study report (CSR), regulatory submissions, and future manuscripts. In addition, post hoc exploratory analyses not necessarily identified in this SAP may be performed to further examine study data. Any post hoc, or unplanned, exploratory analyses performed will be clearly identified as such in the final CSR and in any publications.

Any significant changes from planned analyses will also be described in the final CSR.

Effective: 17/SEP/2020 


#### 3. PROJECT OVERVIEW

### 3.1 Study Design

This is an open-label, adaptive study that will utilise the *P. falciparum* induced blood stage malaria (IBSM) model to characterise the pharmacokinetic/pharmacodynamic (PK/PD) profile and safety of MMV367.

Up to 18 participants will be enrolled in cohorts of up to 6 participants each. The study will proceed as follows for all participants:

- Screening period of up to 28 days to recruit healthy adult participants.
- Day 0: Intravenous inoculation with approximately 2,800 viable *P. falciparum*-infected erythrocytes.
- Days 1-3: Daily follow up via phone call or text message.
- Days 4-7: Daily site visits for clinical evaluation and blood sampling to monitor malaria parasitaemia via quantitative polymerase chain reaction (qPCR).
- Day 7 PM: Start of confinement within the clinical trial unit.
- Day 8: Administration of a single oral dose of the investigational medicinal product (IMP) (MMV367). Different doses of MMV367 will be administered across and within cohorts in order to effectively characterise the PK/PD relationship.
- Days 8-11: Regular clinical evaluation and blood sampling to monitor malaria parasitaemia and measure MMV367 plasma concentration.
- Day 11 AM: End of confinement within clinical trial unit.
- Days 12-23: Outpatient follow-up for clinical evaluation and blood sampling.
- Day 24: Initiation of compulsory definitive antimalarial treatment with Riamet® (artemether/lumefantrine) and/or other registered antimalarials if required. Treatment will be initiated earlier than Day 24 in the event of:
  - Insufficient parasite clearance following IMP dosing (parasitaemia not reduced ≥10fold by Day 10 compared with peak parasitaemia on Day 8).
  - o Parasite regrowth following IMP dosing (initial parasite clearance is followed by asexual parasite regrowth above 5000 parasites/mL).
  - o Participant discontinuation/withdrawal
  - o Investigator's discretion in the interest of participant safety.
- Day 27: End of study visit for final clinical evaluation and to ensure complete clearance of malaria parasitaemia (at least one negative malaria PCR result required).

MMV367 will be administered as a single oral dose on Day 8, with different doses to be tested across and within cohorts to effectively characterise the PK/PD relationship. Participants will be randomised to a dose group on the day of dosing. The highest dose of MMV367 administered in this study will be no more than 1500 mg.

The doses to be tested in Cohort 1 will be as follows:

| MMV367 dose | 20 mg | 90 mg | 1500 mg |
|------------------------|-------|-------|---------|
| Number of participants | 3 | 2 | 1 |


The Safety Data Review Team (SDRT) will meet following the completion of Cohort 1 to review all safety, PK, and PD data. Doses to be tested in Cohort 2 will be informed by the results obtained in Cohort 1 and will be designed to refine the PK/PD parameter estimates. It may be necessary to test a dose lower than 20 mg in Cohort 2 if PK/PD parameters such as the EC50 were not sufficiently well estimated in Cohort 1. It may also be necessary to obtain additional data at the dose levels tested in Cohort 1. The maximum dose in Cohort 2 will not exceed 1500 mg. Specific doses, and the number of participants per dose, to be tested in Cohort 2 will be decided by the SDRT based on PK/PD simulations.

The SDRT will meet following the completion of Cohort 2 to review all safety, PK, and PD data. If the SDRT deems sufficient data has been obtained to achieve the primary endpoint (i.e., the PK/PD relationship of MMV367 has been appropriately characterized), a third cohort of participants will not be enrolled. If the SDRT deems further data is necessary, doses for Cohort 3 will be selected as described above for Cohort 2.

### 3.2 Schema




### 3.3 Schedule of Activities

The below table summarises the activities and procedures to be conducted as per this protocol during screening, eligibility, malaria inoculation, out patient monitoring, IMP administration and clinic confinement, and at the end of study.

# Screening and malaria challenge period

| Study Day | -28 to -1 | -3 to -1 | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 AM |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | Eligibility confirmation | Pre-<br>inoculation | Post-<br>inoculation | Pho | ne cor | ntact | Outpatient visits | | | |
| Informed consent | X | | | | | | | | | | |
| Beck Depression Inventory | X | | | | | | | | | | |
| Cardiovascular risk | Х | | | | | | | | | | |
| Demography | X | | | | | | | | | | |
| Medical history | Х | | Х | | | | | | | | |
| Prior medications | Х | | Х | | | | | | | | |
| Eligibility | Х | X | Х | | | | | | | | |
| Urine drug screen | Х | | X | | | | | | | | |
| Alcohol breath test | X | | Х | | | | | | | | |
| Viral screen blood sample | Х | | | | | | | | | | |
| RBC alloantibody blood sample | Х | | | | | | | | | | |
| Coagulation profile blood sample | Х | | | | | | | | | | |
| COVID-19 rapid test | | | Х | | | | | | | | |
| COVID-19 PCR test | | X | | | | | | | | Х | |
| G6PD test blood sample | Х | | | | | | | | | | |
| Serum pregnancy test blood sample | Xc | Xd | | | | | | | | | |
| Urine pregnancy test (WOCBP) | | | Х | | | | | | | | |
| FSH test (post-menopausal women) | Х | | | | | | | | | | |
| Urinalysis sample | Х | X | | | | | | | | | |
| Adverse events | | | | Х | Х | Х | Х | Х | Х | Х | Х |
| Concomitant medications | | | | Х | Х | Х | Х | Х | Х | Х | Х |
| Safety serum retention | | | Х | | | | | | | | |
| Full physical exam | Xa | | | | | | | | | | |
| Abbreviated physical exam | | | Х | | | | | | | | |
| Symptom directed physical exam | | | | | | | | Х | Х | Х | Х |
| Malaria clinical score | | | Х | | | | | Х | Х | Х | Х |
| Vital signs | Xe | | Х | Х | | | | Х | Х | Х | Х |
| Electrocardiograph (triplicate) | Х | | Х | | | | | | | | |
| Haematology blood sample | Х | X | | | | | | | | | Х |


| Study Day | -28 to -1 | -3 to -1 | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 AM |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Biochemistry blood sample | Xb | X | | | | | | | | | Х |
| Diary card | | | | X | Х | Х | Х | Х | Х | Х | Х |
| Phone contact | | | | | Х | Х | Х | | | | |
| Malaria challenge agent administration | | | | X | | | | | | | |
| Malaria PCR blood sample | | | X | | | | | Х | Х | Χ | Х |
| Future malaria research blood sample (if | | | | | | | | | | | |
| participant consented) | | | ^ | | | | | | | | |

FSH: Follicle-stimulating hormone; G6PD: Glucose-6-phosphate dehydrogenase; PCR: Polymerase chain reaction; RBC: Red blood cell; WOCBP: Women of childbearing potential.


IMP administration and clinic confinement period

| Study Day | 7 PM | • | | | | 8 | | | | | | | 9 | | | 10 | | 11 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Hours post-IMP dose | | Pre-dose | 0 | 1 | 2 | 3 | 4 | 6 | 8 | 12 | 16 | 24 | 30 | 36 | 48 | 54 | 60 | 72 |
| Urine drug screen | Х | | | | | | | | | | | | | | | | | |
| Alcohol breath test | Х | | | | | | | | | | | | | | | | | |
| COVID-19 rapid test | Х | | | | | | | | | | | | | | | | | |
| Urine pregnancy test (WOCBP) | Х | | | | | | | | | | | | | | | | | |
| Adverse events | | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Concomitant medications | | Х | | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Abbreviated physical exam | | Х | | | | | | | | | | | | | | | | |
| Symptom-directed physical exam | | | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Malaria clinical score | | Х | | | | | | Х | | Х | | Х | Х | Х | Х | Χ | Х | Х |
| Vital signs | | Х | | | | | | Х | | Х | | Х | Х | Х | Х | Х | Х | Х |
| Electrocardiograph | | Х | | | | | | | | | | Х | | | Х | | | Х |
| Haematology blood sample | | Х | | | | | | | | | | Х | | | | | | Х |
| Biochemistry blood sample | | Х | | | | | | | | | | Х | | | | | | Х |
| Malaria PCR blood sample | | X | | | Х | | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Randomisation | | Х | | | | | | | | | | | | | | | | |
| IMP administration | | | Х | | | | | | | | | | | | | | | |

<sup>&</sup>lt;sup>a</sup>Body height to be recorded at screening only.

<sup>&</sup>lt;sup>b</sup>Lipids included at Screening for cardiovascular risk factor.

Serum pregnancy test to be performed for all women at Screening.

<sup>&</sup>lt;sup>d</sup>Serum pregnancy test to be performed for WOCBP at the eligibility confirmation visit.

eAt screening, vital signs will be measured after the participant has rested in the supine position for 5 minutes. SBP and DBP will be measured again after the participant has transitioned to a standing position for 3 minutes to assess postural hypotension (see Section 5.2, exclusion criterion 10). At all other time-points vital signs will be measured after the participant has rested in the seated position for at least 5 min.


| IMP PK blood sample | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Χ | Χ | Χ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parasite ex vivo viability blood sample | Х | | | | | | Х | | Х | Х | Х | Х | | Х |
| Future malaria research blood sample (if participant consented)_ | Х | | | | | | | | | | | | | |

IMP: Investigational medicinal product; PK: Pharmacokinetics; PCR: Polymerase chain reaction; WOCBP: Women of childbearing potential.

**Outpatient follow-up period** 

| Study Day | 12 | 13 | 15 | 17 <sup>d</sup> | <b>20</b> <sup>d</sup> | 22 | 24 <sup>d</sup> | 27 EOS <sup>e</sup> |
|---|---|---|---|---|---|---|---|---|
| Hours (days) post-IMP dose | 96±4 (4) | 120±12 (5) | 168±24 (7) | 216±24 (9) | 288±24 (12) | 336±24 (14) | 384±24 (16) | 456±24 (19) |
| Viral screen blood sample | | | | | | | | X |
| RBC alloantibody blood sample | | | | | | | | X |
| Serum pregnancy test blood sample (WOCBP) | | | | | | | | X |
| Urinalysis sample | | | | | | | | X |
| Adverse events | Χ | X | X | X | X | Χ | Χ | Χ |
| Concomitant medications | X | X | X | X | X | X | X | Χ |
| Safety serum retention blood sample | | | | | | | | X |
| Full physical exam | | | | | | | | X |
| Symptom directed physical exam | X | X | X | X | X | X | X | |
| Vital signs | X | X | X | X | X | X | X | X |
| Malaria clinical score | X | X | X | X | X | X | X | X |
| Electrocardiograph | | | | | | | | X |
| Haematology blood sample | | | X | | | X | | X |
| Biochemistry blood sample | | | X | | | X | | X |
| Diary card | X | X | X | X | X | X | X | X |
| Malaria PCR blood sample | X | X | X | X | X | X | X | X |
| IMP PK blood sample | X | X | X | X | X | | | |
| Definitive antimalarial treatment | | | | | | | Xp | |
| Parasite drug resistance blood sample | | | | Xa | | | | |
| Parasite <i>ex vivo</i> growth blood sample | X | | | | Xc | | | |
| Future malaria research blood sample (if participant consented) | Х | | Х | | | | | Х |

EOS: End of study; IMP: Investigational medicinal product; PK: Pharmacokinetics; PCR: Polymerase chain reaction; RBC: Red blood cell; WOCBP: Women of childbearing potential.


<sup>&</sup>lt;sup>a</sup>One blood sample will be collected for parasite drug resistance assessment only in the event of parasite regrowth. This sample will be collected just prior to initiation of definitive antimalarial treatment.

Definitive antimalarial treatment to be initiated on Day 24, or earlier in accordance with the criteria specified in section 4.1 of the protocol.

One blood sample will be collected for parasite ex vivo growth only in the event of parasite regrowth. This sample will be collected just prior to initiation of definitive antimalarial treatment.

<sup>&</sup>lt;sup>d</sup>Visit not required if participant has previously been administered definitive antimalarial treatment and returned at least one negative malaria PCR result.

eParticipants who withdraw, or are withdrawn or discontinued from the trial, will be asked to attend an early termination visit with assessments equivalent to the Day 27 EOS visit.


### 3.4 Objectives

### 3.4.1 Primary Objective

• To characterise the PK/PD relationship of MMV367 in healthy participants experimentally infected with blood stage *P. falciparum*.

### 3.4.2 Secondary Objective(s)

- To evaluate the safety and tolerability of single oral doses of MMV367 in healthy participants experimentally infected with blood stage *P. falciparum*.
- To evaluate the safety and tolerability associated with blood-stage malaria infection in healthy malaria naïve participants.
- To characterise the pharmacokinetics of MMV367 following single oral dose administration in healthy participants experimentally infected with blood stage P. falciparum.
- To characterise the parasite clearance kinetics following single doses of MMV367 in healthy participants experimentally infected with blood-stage *P. falciparum*.

### 3.4.3 Exploratory Objective(s)

- To investigate potential resistance of *P. falciparum* to MMV367 in participants experiencing parasite regrowth after MMV367 administration.
- To characterise the effect of MMV367 on *P. falciparum* parasite viability.

### 3.5 Endpoints

### 3.5.1 Primary Endpoint (s)

• The PK/PD relationship between MMV367 plasma concentrations and blood stage asexual parasitaemia.

### 3.5.2 Secondary Endpoint (s)

### 3.5.2.1 Safety Parameters

- The incidence, severity and relationship to MMV367 of adverse events as determined by self-reported symptoms, clinical laboratory analysis, vital signs, physical examinations and ECG assessments.
- The incidence, severity and relationship to the malaria challenge agent of adverse events as determined by self-reported symptoms, clinical laboratory analysis, vital signs, physical examinations and ECG assessments. Additionally, the severity of the induced malaria infection in each participant graded by the malaria clinical score.

#### 3.5.2.2 PK Parameters

The pharmacokinetics of MMV367 calculated using non-compartmental methods.
 Parameters:

C<sub>max</sub>: Maximum plasma concentration observed

t<sub>max</sub>: Time to reach maximum plasma concentration

AUC<sub>last</sub>: Area under the curve from time 0 to last measurable concentration

AUC<sub>inf</sub>: Area under the curve from time 0 to infinity

t<sub>1/2</sub>: Half-life

CL/F: Apparent Oral Clearance

Effective: 17/SEP/2020 


V<sub>z</sub>/F: Apparent volume of distribution

 $\lambda_{z}$ : Terminal rate constant

#### 3.5.2.3 Parasite Clearance Kinetics

 The parasite clearance kinetics following dosing with MMV367 (parasite reduction ratio over a 48-hour period [PRR<sub>48</sub>] and corresponding parasite clearance half-life [PCt<sub>1/2</sub>]).

### 3.5.3 Exploratory Endpoint (s)

- Incidence and level of resistance to MMV367 in parasites determined using *in vitro* methods.
- The effect of MMV367 on parasite viability examined by ex vivo cultures.

### 3.6 Sample Size

A maximum sample size of up to 18 participants is expected to be sufficient to achieve the primary endpoint of the study, which is to determine the PK/PD parameters of MMV367. This sample size is not based on formal statistical calculations but rather is based on previous experience of characterising the PK/PD relationship of antimalarials using the IBSM model. The specific number of participants required will be dependent on the emerging results during the study; it is possible that less than 18 participants will be required. The SDRT will review the data after the completion of each cohort and decide when sufficient data has been obtained to complete the primary endpoint. No more than 18 participants will be administered IMP in this study.

### 3.7 Treatment Assignment and Randomisation

All participants will receive an identification number (screening number) as soon as they have signed the informed consent form. Participants who meet the eligibility criteria and are enrolled in the study will be assigned an enrolment number on Day 0 immediately prior to administration of the malaria challenge agent. Participants will be randomised within each cohort to a dose group on Day 8, immediately prior to administration of the IMP. A randomisation schedule will be prepared in advance and take in account potential participant withdrawals prior to scheduled dosing with IMP. The details of the randomisation procedure will be described in the randomisation plan. This is an open label study and therefore no blinding will be performed.

### Replacement of Withdrawn/Discontinued Participants

Participants who withdraw, or are withdrawn or discontinued from the trial, may be replaced after mutual agreement between the Sponsor and the Principal Investigator. The decision regarding the replacement of participants will be documented.

All withdrawn participants must successfully complete the full course of definitive antimalarial treatment.

BM S01-A, v3.0

Statistical Analysis Plan


### 4. STATISTICAL CONSIDERATIONS

Data analysis will be performed according to the Sponsor's representative Standard Operating Procedures (SOPs).

The general analytical approach for all endpoints will be descriptive in nature. All summaries will present the data by dose group as well as by all participants combined.

Unless otherwise stated, the following statistical approaches will be taken:

<u>Continuous variables:</u> Descriptive statistics will include the number of non-missing

values, mean, standard deviation (SD), CV%, median,

interquartile range, minimum, and maximum. The minimum and maximum values will be presented to the same number of decimal places as recorded in the raw data; mean and median will be presented to 1 decimal place more than raw data; and SD will be presented to two more decimal places than the raw data. The number of decimals for lab parameters may be reduced if the full presentation of the data includes more than 4

significant figures.

Categorical variables: Descriptive statistics will include frequency counts and

percentages per category. Percentages will be rounded to one decimal place, with the denominator being the number of

patients in the relevant population.

<u>Imputation</u>: No imputation will be performed for missing data.

Confidence intervals (CIs): CIs will be two-sided and will use 95% confidence levels.

Unscheduled Visits Unscheduled visits that do not have laboratory data on the same

visit date will be excluded from summary tables.

<u>Early termination visit</u> Assessments conducted at Early Termination will be excluded

from visit-based summary tables unless otherwise indicated.

### 4.1 Data Capture

#### 4.1.1 Database

The primary method of data collection is via the study database, developed within the chosen Electronic Data Capture (EDC) platform, IBM Clinical Development. The database has been designed based on the final protocol, the system/core configuration, electronic Case Report Form (eCRF) specifications and/or mock eCRF and consistency check specifications.

Data will be entered directly into the EDC system. Site-collected data will be entered directly from source notes at the site and will be verified by Clinical Research Associates (CRAs) to ensure data integrity.

Refer to the Data Management Plan for further details.

### 4.1.2. Third Party Data

### 4.1.2.1 Safety Laboratory

BM S01-A, v3.0

Statistical Analysis Plan Effective: 17/SEP/2020 **CONFIDENTIAL** 


Central safety laboratory data will be received from Sullivan Nicolaides (SNP) Pathology Central Laboratory as specified in the Data Transfer Specification. At least one transfer will be delivered prior to database lock and reconciled against CRF data. Following successful reconciliation and resolution of any data issues, the data will be incorporated into the End of Study analysis.

No unit conversion of laboratory data will be performed.

### 4.1.2.2 PK Laboratory

PK samples will be analysed by Swiss BioQuant Central (SBQ) and PK parameters will be derived by PharmaKinetic. Final PK assay data will be transferred to SSR, as specified in the SBQ DTS, for incorporation into the PC SDTM.

### 4.1.2.3 PD Laboratory

All parasitaemia data will be generated by the Queensland Paediatric Infectious Diseases (QPID) laboratory and captured electronically using MARS (18S qPCR parasitaemia data). All parasite life-stage data (i.e. gametocytemia and ring-stage parasites) will be generated by the QPID laboratory and transferred electronically to the Queensland Institute of Medical Research (QIMR) Berghofer and this data will be used for PK/PD modelling. QIMR will provide the 'raw' PCR data 18S, the female gametocyte-specific transcript (pfs25), the male gametocyte-specific transcript (pfMGET) and the ring-stage transcript (pfSBP-1) to SSR as per DTS, and final PD parameters will be in the PRR report.

### 4.1.2.4 PK/PD Laboratory

PK/PD analysis will be performed by MMV, Pharmacometrics. SSR will be required to provide the PK concentration and parasitemia data, as well as any CRF datasets required to perform the PK/PD analyses (e.g. demographics, drug administration data).

### 4.2 Statistical Programming

### 4.2.1 Programming Specifications

### 4.2.1.1 Safety Analysis

Programming specifications will be prepared to detail the SAS programming of CDISC (SDTM and ADaM) datasets and listings, tables and figures.

#### 4.2.1.2 PD Analysis

Data manipulation and data analyses for all PD data will be performed using R (version 4.1.0 or higher).

### 4.2.1.3 PK Analysis

The estimation of pharmacokinetic parameters by non-compartmental analysis (NCA) methods will be performed using Phoenix WinNonlin software (v8.3 or a more recent version, Certara USA, Inc., USA).

#### 4.2.1.4 PKPD Analysis

All data processing, analysis, model setup and modeling result analysis including goodness-of-fit plots will be performed using R 3.6.3 or above and IQRtools package 1.8.0 or above.

BM S01-A, v3.0


NLME modelling will be performed with Monolix 2019R1 [MLX19] using Stochastic Approximation Expectation Maximization (SAEM) for parameter estimation. For PD modelling where typically the variance of random-effects cannot be estimated from the data, the IQRtools SysFit approach will be used to estimate typical and individual PD parameters.

### 4.2.2 Baseline

Baseline will be defined as:

### Safety

- The last scheduled observation prior to the administration of the malaria challenge inoculum [Inoculation Baseline],
- The last scheduled observation prior to the first administration of IMP [Treatment Baseline].

For replicate measurements (e.g., ECG) at baseline, the mean of those replicates will be used as the baseline value.

### PD

The last observation prior to the administration of the IMP for PD data.

#### PK

• The last observation prior to the administration of the IMP for PK data.

### 4.2.3 Change from Baseline

Change from Baseline will be calculated as:

Change from baseline =  $(postbaseline\ value) - baseline\ value$ 

### 4.2.3.1 Days relative to Inoculation

 $Days = (Assessment \ Date - Inoculation \ Administration \ Date) + 1$ 

### 4.2.3.2 Days relative to IMP administration

 $Days = (Assessment \ Date - First \ Study \ Drug \ Administration \ Date) + 1$ 

### 4.2.4 IMP Treatment Groups

Tabulations will summarise data by the IMP dose groups and these may vary for each cohort.

### 5. ANALYSIS SETS

The analysis sets to be used for the analyses will be: Full Analyses set (FAS), IMP set, PK set, PD set and PK/PD set.

The number of participants in each analysis set will be summarised, with a corresponding listing.

### **5.1 Analysis Set Descriptions**

### 5.1.1 Full Analysis Set

BM S01-A, v3.0

Statistical Analysis Plan Effective: 17/SEP/2020


The Full Analysis Set (FAS) will consist of all enrolled participants, i.e. participants that received the malaria challenge agent.

### 5.1.2 IMP Set

The IMP Set will include all enrolled participants administered with the IMP.

### 5.1.3 PK Analysis Set

The PK analysis set will include all participants who have sufficient plasma samples taken for at least one of the PK parameters to be calculated and who received any study treatment and experienced no protocol deviations with relevant impact on PK data. Should an adverse event, for example, vomiting within 4 hours of IMP dosing occur and be deemed detrimental to the data quality, additional subsets may be invoked, and those participants be omitted from the summary statistics. This will be confirmed by the sponsor if applicable.

### 5.1.4 PD Analysis Set

The PD analysis set will include all participants inoculated with the malaria challenge agent and who develop parasitaemia detectable by qPCR, received a dose of MMV367, and have no protocol deviations that would exclude them from the PD analysis due to their impact on the PD analysis.

### 5.1.5 PK/PD Analysis Set

The PK/PD analysis set will include all participants included in both the PK set and the PD set.

### 6. PROTOCOL DEVIATIONS

Analysis Set: FAS

All protocol deviations will be listed, grouped by participant and dose group.

The protocol deviation summary table will capture all deviations as minor and major.

The protocol deviation summary table will include:

- The total number of minor protocol deviations
- The total number of major protocol deviations
- The number of Participants who reported at least one minor protocol deviation
- The number of Participants who reported at least one major protocol deviation


#### 7. PARTICIPANT DISPOSITION

Analysis Set: FAS

### 7.1 Disposition

A listing of participant disposition will present:

- Date of informed consent
- Date of inoculation
- Date of IMP administration
- Date of mandatory rescue medication administration
- Date of Primacin administration when applicable
- Did the participant complete the study?
- Date of completion / early withdrawal
- Primary reason for early withdrawal (including instances where early termination was related to COVID-19)

Detailed early withdrawal information will also be listed in a separate listing.

If there are any deaths reported, a separate death listing will be prepared.

The number and percentage of Participants entering and discontinuing the study will be summarised by dose group and overall along with the reason for discontinuation. The participant disposition summary table will include:

- Number of participants signed informed consent
- Number of participants who received IMP
- Number of participants who completed the full study
- Number of participants withdrawn from the study early
- Reason for early withdrawal

### 7.2 Analysis of Population Assignment

Analysis set data will be listed for all participants. A summary table will show the number of participants within each of the analysis sets.

#### 8. DEMOGRAPHIC AND BASELINE INFORMATION

Analysis Set: FAS

### 8.1 Demographics

Demographic data will be listed for all enrolled participants and summarised by dose group and overall. Data includes:

Age

Sex

Women of Child-bearing potential

Post-menopausal women

Race

Ethnicity

Weight (kg)

Height (m)

BMI (kg/m<sup>2</sup>)

### 8.2 Medical History

All medical history data will be listed, grouped by participant.

BM S01-A, v3.0

Statistical Analysis Plan Effective: 17/SEP/2020 CONFIDENTIAL


Medical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA version 24.1) and summarised by system organ class (SOC) and preferred term (PT).

#### 8.3 Prior Medications

Prior medications are defined as any medication that is started before first inoculation with the malaria challenge agent, regardless of when it ended. If a medication has a missing or partial missing start/end date or time and it cannot be determined whether it was taken before IMP or concomitantly, it will be considered as prior and concomitant. Medications will be coded using WHODrug Dictionary September 2021 release.

Prior medications will be listed.

### 8.4 Drug Screen

Drug screen data will be listed for all participants.

### 8.5 Alcohol Screen

Alcohol screening data will be listed for all participants.

### 8.6 SARS-CoV-2 Screening

Any positive SARS-CoV2 screening results will be listed.

### 8.7 Follicle Stimulating Hormone (FSH)

FSH results will be listed for Post-menopausal women only.

### 8.8 Beck Depression Inventory

Beck Depression Inventory (BDI-II) data will be listed for all participants, including answers to the individual questions as well as the total scores, which are auto-calculated within the CRF.

BM S01-A, v3.0

Statistical Analysis Plan

Effective: 17/SEP/2020 


#### 9. TREATMENT EXPOSURE

Analysis Set: FAS Set

Participant exposure to the protocol-specified treatments (IMP, malaria challenge agent, mandatory rescue medications - Riamet, Malarone, IV artesunate - and Primacin if also administered) will be listed and summarised by dose of IMP and overall.

### 10. PRIMARY ENDPOINT ANALYSIS (PK/PD ANALYSIS)

Analysis Set: PK/PD Analysis Set

The primary endpoint is the PK/PD relationship of MMV367.

### 10.1 Overview of methodology for PK/ PD Modelling

Two stage approach:

- 1. Estimate the PK parameters by fitting a PK model and relevant covariates to the individual PK concentrations
- 2. Estimate the PD parameters by fitting a PKPD model to the asexual parasitemia observations using the individual PK parameters as regressors

### 10.2 Sources of Data

The PK/PD dataset will contain the individual information on the inoculum volume, date and time of its administration; doses of MMV367 administered with date and time of administration; plasma PK concentrations of MMV367 with date and time of blood sampling; triplicate total parasitemia counts by 18S qPCR with date and time of blood sampling; gametocytemia counts by pfs25, pfMGET and pfSBP-1 if relevant; and typical covariates such as age, body weight, height, sex and race.

The PK/PD dataset will contain the data from the current VIS study MMV\_MMV367\_22\_01 and from the past MMV\_MMV367\_21\_01\_FIH study.

The PK/PD dataset for MMV\_MMV367\_22\_01 will be prepared by SSR in the MMV format from the database. The PK dataset for MMV\_MMV367\_21\_01\_FIH will be prepared by ClinBay.

### 10.3 Data Assembly

#### 10.3.1 Master PK/PD dataset

Data from study MMV\_MMV367\_22\_01\_VIS will contain information on the individual MMV367 doses, MMV367 PK concentrations, the triplicated parasitemia levels, gametocyte data and typical covariates such as age, height, weight, sex and race. Data from study MMV\_MMV367\_21\_01\_FiH will be added to increase the number of individuals with PK profiles.

A master dataset will be assembled formatted according to the MMV dataset standard. (cf., "MS\_IQdataset\_V4"). Plasma concentration will be in ug/mL, total parasite levels in counts/mL, and doses in mg. Gametocyte data is in copies/uL.

Parasite data after the first administration of rescue medication is flagged by setting the IGNORE column to "Rescued". The time in hours is relative to the (first) MMV367 administration time. Gametocyte data will be converted to parasite counts following the

BM S01-A, v3.0


instructions in "Analyzing RNA data by K.Collins Nov2017.docx". Total counts of parasites were flagged to be ignored (by setting the column IGNORE to "gametocytes") if counts of gametocytes exceeded 10% of total counts.

A general analysis dataset will then be created from the master dataset. The general dataset will contain the following observations: MMV367 plasma concentrations, total parasite count, as well as counts of gametocytes. In addition, dosing records for *P. falciparum* inoculation, MMV367 administration and rescue medication administration will be defined.

The following covariates will be included as additional columns in the general dataset.

- DOSELEVEL: the dose amount
- DOSEMULT: the number of doses
- WT0: body weight (kg)
- AGE: age (years)
- SEX: sex (male or female)
- Infection status (for all participants from MMV\_MMV367\_22\_01\_VIS infection status will be positive; For all participants from MMV\_MMV367\_21\_01\_FIH infection status will be negative.)
- PLbase: The model baseline parasitemia value the geometric mean of parasite counts at time of first MMV367 dose.

### 10.3.2 PK modeling data set

Observations below the lower limit of quantification (LLOQ) will be censored by setting the CENS column for these observation records to 1 and setting the corresponding dependent variable (DV) column to the LLOQ (→ M4 method). Observation records with missing values and records with missing times will be ignored. Records flagged to be ignored will be removed from the dataset. Observations not analyzed in the PK modelling (i.e., all parasite count records) will be removed. Consequently, the PK modelling NLME dataset will contain only MMV367 dosing records and MMV367 plasma concentration records.

### 10.3.3 PD modeling data set

Observations below the LLOQ will be censored by setting the CENS column for these observation records to 1 and the corresponding DV value to the LLOQ, i.e., 10 p/mL ( $\rightarrow$  M3 method). Total and viable counts of parasites for which counts of gametocytes exceeded 10% of total counts are flagged to be ignored (by setting the column IGNORE to "gametocytes"). Observation records with missing values and records with missing times will be ignored. Records flagged to be ignored will be removed from the dataset. Observations not analysed in the PD modelling analysis (i.e., MMV367 plasma concentration records) will be removed. Consequently, the PD modelling NLME dataset will contain only MMV367 dosing records and total parasite counts.

Parasite counts will be log-transformed for the PD modelling and estimated individual PK model parameters will be added to the dataset as regressors.


#### 10.4. Methods

### 10.4.1. General PKPD model building approach

Population models of the PK and PD will be developed in step-wise manner.

BM S01-A, v3.0


1. A population PK model will be developed to obtain individual PK parameter estimates based on which the individual PK profiles are well described.

- 2. A parasite growth model (parasite growth rate and deviation of parasitemia at inoculation from parasitemia at IMP administration) will be estimated from the total parasite counts before treatment administration. Estimation of typical and individual PD parameters will be performed with IQRtools SysFit. Other appropriate growth models, e.g. an oscillatory model, will be tested if advisable.
- 3. The PKPD model will be built using the individual PK parameter estimates and individual growth model parameter estimates as regression parameters. Estimation of typical and individual PD parameters will first be performed with IQRtools SysFit to investigate model identifiability and second with Monolix to additionally estimate IIV.

Estimations will be done using gradient-based SysFit algorithm in IQRtools or SAEM algorithm in Monolix. Other appropriate methods may be used if advisable.

Inter-individual variability (IIV) is implemented for normally distributed parameters using the following equation with  $\theta_0$  as population average parameter,  $\theta_i$  as individual parameter, and  $\eta_i$  as random effect that is distributed normally around zero  $(\eta_i \sim N(0, \omega^2))$ .

$$\Theta_i = \Theta_0 + \eta_i$$

The following equation is used for log-normally distributed parameters.

$$\ln(\theta_i) = \ln(\theta_0) + \eta_i$$

Continuous covariates on log-normally distributed parameters will be implemented as follows.

$$\Theta_i = \Theta_0 \cdot \frac{COV_i}{COV_{median}}^{\beta} \cdot e^{\eta_i}$$

 $\Theta_i$  represents the individual parameter,  $\Theta_0$  the population mean value,  $COV_i$  the individual covariate value,  $COV_{median}$ , the population median covariate value,  $\beta$  the covariate coefficient, and  $\eta_i$  the individual random effect.

Categorical covariates on log-normally distributed parameters will be implemented as follows.

$$\Theta_i = \Theta_0 \cdot \Sigma_i (e^{\beta_j \cdot COV_{ij}}) \cdot e^{\eta_i}$$

The individual covariate values  $COV_{ij}$  are 1 if participant i belongs to the  $j_{th}$  category of the covariate and 0 otherwise.  $beta_j$  is the covariate value for the  $j_{th}$  category. For one category, i.e. the reference,  $beta_i$  is 0.

For the NLME modeling with Monolix, the log-likelihood and the Fisher information matrix will be approximated by importance sampling and stochastic approximation respectively. The number of iterations in the burn-in and the accumulation phase will be 500 and 200 respectively, but might be adjusted if required based on inspection of parameter estimate and objective function traces along estimation iterations. Individual parameters will be determined as conditional modes.

For PD modelling with the IQRtools SysFit implementation, a non-linear fixed-effects modelling approach is employed. Typical and individual parameters are both treated as fixed effects. The parameterization of individual parameters and covariates is fully consistent with the NLME parameterization above. The variances  $\omega^2$  of NLME random effects are accounted for by quadratic priors, added to the log-likelihood function, where the values for  $\omega^2$  are fixed and the  $\eta$  parameters are estimated. The profile-likelihood method [4, 5] is used to compute confidence intervals of the parameters estimated with the SysFit approach.


#### 10.4.1.1. Model evaluation

Assessment of model adequacy and decisions about increasing model complexity will be driven by the data and guided by goodness-of-fit criteria, including:

- visual inspection of diagnostic scatter plots (observed vs. predicted concentration, residual/weighted residual vs. predicted concentration or time and histograms of individual random effects, for example),
- 2. successful convergence of the minimization routine with at least 2 significant digits in parameter estimates,
- 3. plausibility of parameter estimates,
- 4. precision of parameter estimates,
- correlation between model parameter estimation errors<0.95, and 5.
- the Bayesian information criterion (BIC), given the minimum objective function value and number of estimated parameters.

For the nonlinear fixed effects models, additional diagnostic plots will be produced:

- objective function values across multiple fits from randomised initial guesses, and
- 8. profile likelihood plots

All parameter estimates will be reported with a measure of estimation uncertainty, such as the relative standard error of the estimates. The individual PK fits will be used to evaluate the adequacy to use the individual PK parameter estimates as regression parameters for PD modelina.

The adequacy of simulation with the selected models will be evaluated by visual predictive checks (VPCs). VPCs for each dose level will be performed by simulation of the study 200 times taking parameter estimation uncertainty into account. 95%-confidence intervals for the 5th percentile, the median, and the 95th percentile will be derived and compared to the corresponding values based on the data.

#### 10.4.2. Building a PK model

The PK of MMV367 will be modeled using compartmental models describing the absorption after oral administration, distribution between central and peripheral compartments, and the elimination from the central compartment. The visual data analysis will guide the selection of models that will be tested (e.g., with respect to number of compartments, linear or saturable elimination, absorption kinetics and error model). Covariates will be included if appropriate. Estimations will be done using SAEM algorithm in Monolix. Other appropriate methods may be used if advisable.

FIH data from MMV MMV367 21 01 FIH has previously indicated that MMV367 PK is adequately described by a one-compartment model with first order absorption parameterized in terms of CL/F. Vc/F and ka. Therefore, this structural model will initially be used to model MMV367 PK using the PK modeling dataset. If required to adequately describe MMV367 PK, structural models with greater numbers of compartments and different absorption models (eq first-order rate, lag, transit compartments) will be fitted.

An exploratory investigation of covariate-parameter relationships will be undertaken during the PK modelling step. The covariate WT0 on the clearance and volume parameters will be included to allow predictions in children. Since the body weight distribution may be narrow, the exponents will be fixed to 0.75 and 1 respectively on clearances and volumes of distribution. Other covariates of interest may include AGE, SEX, Infection status and PLbase - however, depending on the population make-up of these covariates, some may not be included. In the event that the distributions of WT0 and AGE are very narrow, a reference value for the population may be used instead of individual participant covariates.

BM S01-A, v3.0

Statistical Analysis Plan


Covariate modeling will be undertaken in the following steps:

- Pre-defined covariate-parameter relationships will be identified based on exploratory analysis and mechanistic plausibility – in particular, WT0 on clearance and volume PK parameters (central and peripheral compartments, if appropriate).
- A full model will be constructed, avoiding simultaneous inclusion of covariates with correlation coefficients >0.5.
- Population parameters will be estimated (both fixed effects [covariate coefficients and structural model parameters] and random effects).
- An exploratory assessment of any remaining trends will be conducted by graphical inspection of all covariate effects (plots of MAP Bayes estimates of individual random effects and/or WRES from the full model vs. covariates).
- Inferences about clinical relevance of parameters will be based on the resulting parameter estimates of the full model and measures of estimation precision (asymptotic standard errors, bootstrap 95% confidence intervals or log-likelihood profile).
- No hypothesis testing will be conducted.
- This approach enables the direct assessment of clinical relevance of covariate effects and also provides some explanation for the apparent absence of a covariate effect (true lack of an effect vs. lack of information about that effect).

Based on diagnostics plot (if shrinkage is less than >30%) the estimation of random effect covariance matrix will be considered. Additionally, it will be attempted to estimate the full random effect covariance matrix. In order to assess the identifiability of the correlations between random effects, parameter estimations will be repeated from randomly chosen initial guesses for the fixed effect parameters that are estimated. All resulting parameters, including the correlation estimates for the random effects will be compared.

### 10.4.3. Building a PD model

PD model development will be done using gradient based algorithms in IQRTools SysFit. The selected model will then be estimated with SAEM in Monolix to attempt to estimate IIV. Other appropriate methods may be used if advisable. As a general concept the changes in living parasite P are modeled as the effect of a net exponential growth rate GR and a killing or clearance rate Kill due to MMV367. The initial parasitemia  $P_{base}$  at time  $t_0$  will be derived from the mean parasitemia which was observed at treatment administration and a parameter PLerr to allow for population and individual deviations. The equations are expressed in the log-scale such as:

$$\frac{dPL}{dt} = GR - Kill$$

$$PL(t_0) = PL_{base} + PLerr$$

where  $PL = \ln(P)$  is the log-transformed parasite counts.

Different models describing the relationship of *MMV367* plasma concentration on the killing rate may be tested.

### 10.5. PK/PD Endpoints

- PK/PD equations comprising the final structural model
- Primary PK and PD parameters that make up the final structural model: estimated typical values with 90% confidence interval

BM S01-A, v3.0


#### 10.6. Presentation of Results

A statistical and graphical analysis of the data (based on the general analysis dataset) will be included.

The analysis results will be reported in the main body of the CSR and technical details will be reported as an appendix (referred to here as the 'technical appendix'). The technical appendix will include the clinical data used in the analysis, data assembly, modelling methods, all results, discussions, and conclusions.

Key results will include description and interpretation of the selected model, parameter estimates, diagnostic plots of goodness-of-fit and will be included in the main text. Limitations of the model prediction will be discussed in the Discussion section of the technical appendix and mentioned in the main text of the CSR.

### 11. SECONDARY ENDPOINTS ANALYSIS

### 11.1 PD Analysis

Analysis Set: PD Analysis Set

PD endpoint: The parasite clearance kinetics following dosing with MMV367.

### 11.1.1 Data Handling

### Handling of replicates

The data will be recorded as triplicate parasitaemia values for each participant at each time point. The replicate data will be summarised by calculating the geometric mean of the parasitaemia values per participant and time point and will be log10 transformed for statistical analyses.

#### Handling of missing data

Missing parasitaemia data will not be imputed. For any replicates that were non-detects (ND), the value will be substituted with 1 parasite/mL prior to calculating the geometric mean for parasitemia quantified from qPCR.

#### 11.1.2 Parasite clearance kinetics

The Parasite Reduction Ratio (PRR) and corresponding parasite clearance half-life (PCt $_{1/2}$ ) of asexual parasites is derived from the clearance rate of parasitaemia after administration of MMV367 treatment. The analysis of PD response to investigational antimalarial therapy consists of:

- calculating the optimal parasite clearance rate (slope coefficient from the log-linear decay regression of qPCR data) for each individual, then,
- estimating dose specific parasite clearance rate and 95% confidence interval (CI) by calculating the weighted average slope estimate and corresponding standard error (SE) using an inverse-variance method.

The data used for all model selection and fitting calculations is comprised of the log<sub>10</sub> transformed geometric mean of parasitaemia per time point per participant up to the first time point all parasitaemia replicates are ND. If during initial parasite clearance there are no samples ND for a participant, the last time point included in the analyses will be three time points after the minimum observed parasitemia value. All subsequent time points are set to 'missing' regardless of whether parasitaemia values increased afterwards due to potential

BM S01-A, v3.0

Statistical Analysis Plan

Effective: 17/SEP/2020 


recrudescence. Sensitivity analyses may be performed using other thresholds to determine parasite clearance, for example, but not limited to, the lower limit of quantification (LOQ) (i.e. the lower limit of the reportable range) of 32 parasites/mL or limit of detection of 111 parasites/mL [1], to assess robustness of PRR estimates.

The PRR per 48 hours, PRR<sub>48</sub>, for asexual parasite will be estimated using the slope of the optimal fit of the log-linear relationship of the parasitaemia decay over time from MMV367 administration for each individual, as detailed in CTM QIMR SOP 41 and Marquart et al. [2]

Table 1: Symbols and definitions of terms used in parasite clearance analysis (Part 1)

| Symbol | Definition |
|---|---|
| PRR <sub>48,i</sub> | Individual specific Parasite Reduction Ratio per 48 h |
| PRR <sub>48,D</sub> | Dose specific Parasite Reduction Ratio per 48 h |
| $\beta_{1,i}$ | Slope coefficient of log10 parasitaemia vs. time profile for individual <i>i</i> |
| $SE_{\beta_{1,i}}$ | SE corresponding to $eta_{1,i}$ for individual $i$ |
| $ar{eta}_{1,D}$ | Dose specific average slope estimate |
| $SE(\bar{\beta}_{1,D})$ | Weighted SE of dose specific average slope estimate |
| PCt½ | Parasite clearance half-life |

### Regression Modelling to Determine Optimal Fit

A regression modelling approach to remove potential lag and/or tail phases of the parasitaemia decay profile will be used to determine the optimal log-linear decay regression. The algorithm considers removing parasitaemia data points in an iterative process from both ends of the parasitaemia curve, i.e. a combination of right censoring (removing values from the tail phase) and left censoring (removing values from the lag phase), and uses model selection techniques to find the optimal log-linear regression.

The algorithm to obtain the log-linear decay for each participant is based on the log-linear regression detailed in Equation (1), where Time is the number of hours since administration of antimalarial treatment (Time = 1, ..., m), and  $\beta_0$  and  $\beta_1$  are the intercept and slope estimates, respectively.

$$\log_{10} Parasitemia = \beta_0 + \beta_1 Time \quad (1)$$

Based on the parasitaemia data for each participant, the iterative algorithm to determine the optimal log-linear decay for each participant is summarised in Table 2. The iterative algorithm is continued until a minimum of four observations are available.

The optimal log-linear regression model for a participant is deemed an appropriate fit if the overall model p-value < 0.001.

Table 2: Iteration process to determine the optimal log-linear decay curve.


Step 1: For each participant, fit the full model - fit a linear regression (as defined by Equation 1) to all m parasitaemia values of participant i

Step 2: Fit two models:

- Fit linear regression model to m-1 parasitaemia values, removing the first (a) observation.
- Fit linear regression model to m-1 parasitaemia values, removing the last (b) observation.

Step 3: Determine the best model of Step 2(a) and Step 2(b), defined as the model corresponding to the minimum overall model p-value.

Step 4: Of the best model defined in Step 3, repeat Step 2 and Step 3 in an iterative process until a minimum of four observations.

Step 5: Of the m-3 best models selected per iteration (including the full model (Step 1)), the optimal model was defined by the minimum overall model p-value.

### Estimating Participant Specific PRR

The slope and corresponding SE estimate of the optimal linear regression model is used to calculate the participant specific PRR<sub>48</sub> estimate and corresponding 95% confidence interval (95% CI), as shown in Equation (2) and (3), respectively.

$$PRR_{48.i} = 10^{-48 \times \beta_{1,i}} \tag{2}$$

$$PRR_{48,i} = 10^{-48 \times \beta_{1,i}}$$
 (2)  
95% CI:  $10^{-48 \left(\beta_{1,i} \pm 1.96 \times SE(\beta_{1,i})\right)}$  (3)

where  $eta_{1,i}$  and  $SE_{eta(1,i)}$  are the slope and corresponding standard error of the slope parameter of the optimal linear regression model, respectively.

### Estimating Dose Specific PRR (PRR<sub>48.D</sub>)

Of the participants with appropriate overall fit (p<0.001), the average PRR<sub>48</sub> and corresponding 95% CI for each cohort is estimated by using the inverse variance method to calculate the weighted average linear regression slope  $(\overline{\beta_1})$  and corresponding SE. The weighted average slope for s participants in the dose with appropriate overall fit is given by Equation (4):

$$\overline{\beta_1} = \frac{\sum_{i=1}^{S} (w_i \times \beta_{1,i})}{\sum_{i=1}^{n} w_i}, \ i = 1, ..., s$$
 (4)

where the weight is the inverse of the squared standard error,  $w_i = \frac{1}{SE(\beta_{+})^2}$ . The standard

error of 
$$\overline{\beta_1}$$
 is estimated as,  $SE\left(\overline{\beta_1}\right) = \sqrt{\frac{1}{\sum_{i=1}^S w_i}}$  .

Therefore the dose specific PRR (PRR<sub>48.D</sub>) and corresponding 95% confidence interval is estimated as shown in Equation (5) and (6), respectively:

$$PRR_{48,D} = 10^{-48 \times \overline{\beta_1}}$$

$$95\% CI: 10^{-48 \times \left(\overline{\beta_1} \pm 1.96 \times SE(\overline{\beta_1})\right)}$$
(6)

95% 
$$CI$$
:  $10^{-48 \times \left(\overline{\beta_1} \pm 1.96 \times SE(\overline{\beta_1})\right)}$  (6)

PRR<sub>48</sub> estimates will also be reported as log<sub>10</sub>(PRR<sub>48</sub>).

### Parasite Clearance Half Life


The parasite clearance half–life (PCt½) will be derived from the optimal decay rate, as shown in Equation (7):

$$PCt_{1/2} = \frac{\log_{10}(2)}{-\beta_1} \qquad (7)$$

The relationship between PRR<sub>48</sub> and parasite clearance half-life ( $PCt\frac{1}{2}$ ) is a simple transformation of the PRR<sub>48</sub> as shown in Equation (8):

$$PCt_{\frac{1}{2}} = log_{10}(2) \times \left(\frac{48 \ hours}{log_{10}(PRR_{48,i})}\right) = \frac{log_{10}(2)}{-\beta_{1,i}}$$
 (8)

where PRR<sub>48,i</sub> is the parasitaemia ratio estimated over a 48-hour interval that is subsequently transformed into a per hour clearance rate.

## Comparison of Dose Specific PRR<sub>48</sub>

To determine whether there are differences between dose specific PRRs, an omnibus test for between group differences is used. The test is used to assess whether there are differences in the weighted mean slope of the *J* doses, using the test statistic shown in Equation (9),

$$Q_B = \sum_{j=1}^{J} w_j \cdot (\bar{\beta}_j - \bar{\beta}_{..})^2 \sim \chi_{J-1}^2 \qquad j = 1, ..., J \qquad (9)$$

The weight for the  $j^{th}$  dose is denoted by  $w_j = \sum_{i=1}^{s_j} w_{ij}$  for participant i with appropriate overall fit in dose j. The  $\bar{\beta}_j$  is the weighted average slope for dose j as defined in Equation (10), and  $\bar{\beta}_{...}$  is the weighted grand mean given by:

$$\bar{\beta}_{\cdot \cdot} = \frac{\sum_{j=1}^{J} w_{j \cdot} \bar{\beta}_{j \cdot}}{\sum_{j=1}^{J} w_{j \cdot}} \tag{10}$$

Post-hoc pair-wise comparisons can be calculated using the test statistic  $Z_G = \frac{G}{\sqrt{v_G}}$ , where G is the contrast  $(G = c_1 \bar{\beta}_1. + \dots + c_J \bar{\beta}_J)$  and  $v_G$  is the variance of the contrast  $(v_G = \frac{c_1^2}{w_1} + \dots + \frac{c_J^2}{w_J})$ . The p-value of the L pair-wise comparisons can be calculated using the Scheffe method, by comparing  $Z_G^2$  to a chi-squared distribution with L-1 degrees of freedom.

### 11.1.3 Presentation of Results

Parasitaemia data will be listed for all enrolled participants and summarised for the PD population. PD parameters will be presented for all participants included in the PD population.

Parasite life-stage data (pfs25, pfMGET and sbp1 qRT-PCR) will be listed by participant and timepoint.

A full report on the pharmacodynamic data analysis will be included in the appendices of the CSR. This report will include a listing of PD endpoints (PRR<sub>48</sub>, PC<sub>t1/2</sub>), a table for Summary of PD endpoints by dose group and a figure for individual log-parasitaemia regression fit.


List of planned tables, listings and figures are in Appendix, Table A.


#### 11.2 **PK Analysis**

Analysis Set: PK Analysis Set

PK endpoint: The pharmacokinetics of MMV367 calculated using non-compartmental methods.

### 11.2.1 Data Handling

### Imputation of Non-Numerical or Negative Values

The imputation of non-numerical or negative values reported in the input data set will be performed as follows:

- Pre-dose sample times will be entered as zero
- Values that are below the limit of quantification (BLQ) obtained prior to the C<sub>max</sub> will be entered as zero
- Values that are BLQ after the C<sub>max</sub> will be treated as missing.
- Should partial AUCs be required then values that are BLQ after C<sub>max</sub> may be imputed as zero for these partial areas if lambda-z cannot be determined.
- Values that are quantifiable after at least 2 consecutive BLQ values after C<sub>max</sub> will be treated as missing for the calculation of PK parameters.

### Missing data

• Values that are reported as "No Result" or "No Sample" etc. will be treated as missing

### 11.2.2 Rules for Pharmacokinetic Parameter Estimation using WinNonlin

Plasma concentration vs time profiles of MMV367 will be generated for each participant to allow for PK analysis. Pharmacokinetic parameters will be estimated using standard Phoenix WinNonlin methods, details of which may be found in the documentation accompanying the WinNonlin software package. The following constraints will apply:

| Parameter Estimation | Constraint |
|---|---|
| Trapezoidal Method | Linear trapezoidal linear/log interpolation method |
| Number of Points used for Lambda-z | At least 3, not including C <sub>max</sub> |
| Minimum Requirements for AUC | At least 3 consecutive quantifiable concentrations |
| Dose | Actual dose |
| Sampling Times | Actual sampling times |

Where possible, the elimination rate constant (lambda-z) will be calculated for all participants. The value of lambda-z will be determined by the slope of the regression line of the natural log transformed concentrations vs time.

The choice of data points for determination of lambda-z will be applied by the Phoenix software as a default method, the pharmacokineticist who may adjust the selection to provide a more appropriate fit and records of this will be documented in the software data.


### 11.2.3 Data Quality

The following flags/footnotes may be applied to the pharmacokinetic parameters:

BM S01-A, v3.0


| Flag | Footnote |
|---|---|
| а | Rsq of regression was <0.8 |
| b | Extrapolated portion of AUC <sub>0-inf</sub> >20% |
| С | Insufficient post-C <sub>max</sub> data points for estimation of lambda-z |
| d | Entire profile BLQ, no pharmacokinetic parameters could be calculated |
| е | Regression could not be fitted |

In the event that a reliable lambda-z cannot be determined, or the extrapolated portion of  $AUC_{0-inf}$  is >20%, then the parameter estimates derived using lambda-z and/or  $AUC_{0-inf}$  may be deemed unreliable and excluded from the summary statistics. Additional flags may be applied based on emerging data.

### 11.2.4 PK parameters

The following pharmacokinetic parameters for MMV367 in plasma will be estimated where possible and appropriate for each participant and dose group:

| CDISC<br>Term | Parameter | Definition | DP or SF | No. of<br>DP/SF |
|---|---|---|---|---|
| TMAX | $T_{max}$ | Time of maximum observed concentration | DP | 2 |
| CMAX | C <sub>max</sub> | Maximum observed concentration | SF | 3 |
| AUCLST | $\mathrm{AUC}_{\mathrm{last}}$ | Area under the curve from 0 time to the last measurable concentration | SF | 3 |
| AUCIFO | $\mathrm{AUC}_{0	ext{-inf}}$ | Area under the curve from 0 time extrapolated to infinity | SF | 3 |
| LAMZHL | t <sub>1/2</sub> | Apparent elimination half-life | DP | 2 |
| LAMZ | Lambda-z | Slope of the apparent elimination phase | DP | 4 |
| CLFO | CL/F | Total body clearance after extravascular administration | SF | 3 |
| VZFO | V <sub>z</sub> /F | Apparent volume of distribution based on the terminal phase after extravascular administration | SF | 3 |

DP=decimal places SF=significant figures

### 11.2.5 Presentation of Results

All bioanalytical data will be listed and summarised according to the actual sampling timepoint.

If the actual sampling time is not within  $\pm$  20% of the scheduled sampling time, the concentration value at the sampling time point may be excluded from descriptive statistics and PK parameter estimation.

Effective: 17/SEP/2020 


All pharmacokinetic parameters generated will be listed and summarised. Where pharmacokinetic data fails to meet the defined criteria in Section 11.2.3. (Data Quality) the affected results will be excluded from the descriptive statistics will be flagged as per exclusion reason.

### 11.2.5.1. Bioanalytical and PK Parameters Listings

All bioanalytical and pharmacokinetic data generated will be listed in individual tables according to the analyte and treatment.

### 11.2.5.2. Bioanalytical and Pharmacokinetic Summary Tables

Bioanalytical and PK parameters summary tables will be performed by SSR.

Summary statistics (i.e., mean, median, SD, CV%, minimum, maximum, n, geometric mean, geometric SD and geometric CV%) will be calculated for PK results for each time point, parameter and dose group.

All summary statistics (i.e., mean, median, SD, CV%, minimum, maximum and n) will be presented for all PK parameters by dose level. Also, geometric mean, geometric SD and geometric CV% will be presented for all PK parameters (except  $T_{max}$ ) by dose group. The  $T_{max}$  summary statistics will be provided as n, minimum, median, and maximum only.

Additional summary tables might be produced if required and requested.

### 11.2.5.3. Bioanalytical and Pharmacokinetic Figures

All arithmetical mean plasma concentration vs. time curves will be produced by dose group on both linear/linear and  $log_{10}/linear$  scales.

All spaghetti plots of individual plasma concentrations against actual sampling times after dosing grouped by dose level will be produced on both a linear/linear and log<sub>10</sub>/linear scale. Each participant's concentration profile will be represented on these plots with a different symbol and a legend will be included on the plots to define the symbols used.

List of summary tables, listings and figures are in Appendix, Table A.

### 11.3 Safety

Analysis Set: Safety data will use both FAS and IMP Sets

Endpoint: The incidence, severity and relationship to MMV367 and malaria challenge of adverse events.

Safety and tolerability will be assessed by clinical review of the following parameters:

- Adverse events (AEs)
- Vital signs
- 12-lead ECG
- Clinical Laboratory analysis
- · Physical examination

#### 11.3.1. Adverse Events

AEs will be reported according to the volunteer infection studies (VIS) plausible windows and reporting rules:


BM S01-A, v3.0


- Inoculum-emergent AEs (IEAEs)= AEs beginning any time from inoculation with the challenge agent until the end of study.
- Treatment-emergent AEs (TEAEs)= AEs beginning any time from administration of the IMP until the end of study.

Adverse Events of Special Interest (AESIs) may be serious or non-serious and are defined by the Sponsor as being of specific scientific and/or medical concern to the Sponsor's product or program. Evaluation on AESI will be based on both Safety Set and FAS depending on if it is treatment emergent or inoculum emergent adverse events.

Any abnormalities listed below should be reported as an AESI.

### **Hepatic:**

- ALT or AST > 5× ULN
- ALP > 2 × ULN (in the absence of known bone pathology)
- Total bilirubin > 2× ULN (in the absence of known Gilbert syndrome)
- Any AST or ALT value > 2× ULN and total bilirubin > 1.5× ULN
- Any ALT or AST value > 2 × ULN and INR > 1.5
- Potential Hy's Law cases (defined as ALT or AST > 3 × ULN and total bilirubin > 2× ULN [mainly conjugated fraction] without notable increase in ALP to > 2× ULN)
- Any clinical event of jaundice (or equivalent term)
- ALT or AST > 2× ULN accompanied by (general) malaise, fatigue, abdominal pain, nausea, or vomiting, or rash with eosinophilia (eosinophil percent or count above the ULN).

### Cardiac:

- QTcF at any time >480 msec
- Bundle branch block (except right bundle branch block that was present prior to MMV367 administration)
- Any arrhythmia, except:
  - sinus bradycardia that is clinically asymptomatic and not associated with any other relevant ECG abnormalities
  - sinus tachycardia that is clinically asymptomatic, is associated with a body temperature
     >38.0°C, and not associated with any other relevant ECG abnormalities
  - respiratory sinus arrhythmia
  - o wandering atrial pacemaker, or
  - isolated single premature atrial/ventricular complex (i.e., no bigeminy, trigeminy, couplets, triplets or salvos) that does not occur more than once in a particular ECG tracing.

### Haematological:

- Haemoglobin drop >20.0 g/L from baseline (at eligibility visit)
- Absolute neutrophil count (ANC) <0.5 × 10<sup>9</sup>/L.
- Platelet count <75 × 10<sup>9</sup>/L.

### Dermatological: \*†

BM S01-A, v3.0

Statistical Analysis Plan Effective: 17/SEP/2020


Clinical signs of possible cutaneous adverse reactions such as:

- Dermatitis
- Rash including
  - erythematous
  - o macular
  - o papular
  - o maculopapular
  - o pruritic
  - o pustular
  - o vesicular

\*If one of these cutaneous reactions is observed, pictures of the lesions should be obtained when feasible.

†Dermatological AEs need not be reported as AESIs if clearly unrelated to the malaria challenge agent or IMP (e.g. rash from cannula dressing or ECG dots).

### 11.3.1.1. **Parameters**

Parameters to be included in the listings? will be:

- Event Term
- Dates, times and study days of onset and resolution
- Severity (CTCAE Grades 1 to 5)
- Outcome (Not Recovered / Not Resolved; Recovered / Resolved; Recovered / Resolved with Sequelae; Recovering / Resolving; Fatal; Unknown)
- Relationship of AE to IMP (Not Related/Not Suspected, Related/Suspected)
- Relationship of AE to rescue medication (Not Related/Not Suspected, Related/Suspected)
- Relationship of AE to malaria challenge agent (Not Related/Not Suspected, Related/Suspected)
- Relationship of AE to study procedures (Not Related/Not Suspected, Related/Suspected)
- Action taken with IMP (No action taken; Rescue medication administered instead of IMP)
- Other actions taken (including withdrawal from the study)
- Seriousness (and Serious Adverse Event (SAE) criteria)
- AESI status (Yes/No)
- Relatedness to COVID-19 (Yes/No)

Derived parameters:

- Duration in hours
- Time in days of onset relative to first IMP administration

### 11.3.1.2. Biostatistical Methods

All pre-dose AEs occurring before inoculation will be reported as Medical History.

Adverse events (AE) will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA) version 24.1 – Sep 2021 and grouped by system organ class (SOC) and preferred terms (PT). Their severity will be graded according to NCI-CTCAE v5.0 27 Nov 2017.

### 11.3.1.2.1. Listings

All AE data will be listed for each participant, including severity, relationship to IMP, relationship to study procedures, relationship to rescue mediation, relationship to malaria

BM S01-A, v3.0

Statistical Analysis Plan Effective: 17/SEP/2020


challenge agent, outcome and actions taken. In addition, listings of AEs leading to discontinuation of the study, SAEs and deaths, will be provided as applicable.

#### 11.3.1.2.2. **Tables**

The number of events, as well as the number and percentage of participants experiencing an AE, will be summarised by, dose group and overall as follows:

Overall summary of IEAEs (FA set) Overall summary of TEAEs (IMP set)

Summary of IEAEs by System Organ Class and Preferred Term - All Causalities (FA set) Summary of TEAEs by System Organ Class and Preferred Term - All Causalities (IMP set)

Summary of IEAEs by System Organ Class, Preferred Term and Maximum Severity - All Causalities (FA set)

Summary of TEAEs by System Organ Class, Preferred Term and Maximum Severity - All Causalities (IMP set)

Summary of Malaria-Related IEAEs by System Organ Class and Preferred Term (FA set) Summary of IMP-Related TEAEs by System Organ Class and Preferred Term (IMP set)

Summary of Malaria-Related IEAEs by System Organ Class, Preferred Term and Maximum Severity (FA set)

Summary of IMP-Related TEAEs by System Organ Class, Preferred Term and Maximum Severity (IMP set)

Summary of IE SAEs by System Organ Class and Preferred Term - All Causalities (FA set) Summary of TE SAEs by System Organ Class and Preferred Term - All Causalities (IMP set)

Overall Summary of IE AESIs (FA set) Overall Summary of TE AESIs (IMP set)

Summary of IE AESIs by System Organ Class and Preferred Term - All Causalities (FA set) Summary of TE AESIs by System Organ Class and Preferred Term - All Causalities (IMP set

Summary of IEAEs Leading to Study Discontinuation by System Organ Class and Preferred Term - All Causalities (FA set)

Summary of TEAEs Leading to Study Discontinuation by System Organ Class and Preferred Term - All Causalities (IMP set)

For the summary tables, participants who experience the same AE (in terms of the MedDRA preferred term) more than once will only be counted once.


#### 11.3.2. Concomitant Medication

Medications used in this study will be coded using WHODrug Global version B3 Sep 2021 – Added Context.

Concomitant medications are defined as medications continued or newly received at or after administration of the malaria challenge agent through to the End of Study visit.

If a medication has a missing or partial missing start/end date or time and it cannot be determined whether it was taken before initial treatment or concomitantly, it will be considered as prior and concomitant.

Concomitant medications will be summarised by ATC and PN. The summary tables will show the number and percentage of participants taking each medication by ATC and PN.

For the summaries of concomitant medications, participants who take the same medication (in terms of the ATC and PN) more than once will only be counted once for that medication.

Use of rescue medications will be analysed as part of the treatment exposure analysis (Section 9).

BM S01-A, v3.0

Statistical Analysis Plan

Effective: 17/SEP/2020 


### 11.3.3. Laboratory

### **Parameters**

# <u>Haematology</u>

White cell count (WCC)
Neutrophils (NEUT)
Lymphocytes (LYM)
Monocytes (MON)
Eosinophils (EOS)
Basophils (BAS)
Mean cell volume (MCV)
Red cell count (RCC)
Haemoglobin (HGB)
Haematocrit (HCT)
Platelet count (PLAT)
Red cell distribution width (RDW)
Reticulocyte count (RETI)
Blood Group and Rh(D) tests (*Screening only*)

### **Biochemistry**

| Potassium (K) Chloride (CL) Bicarbonate (BICARB) Calcium (CA) Corrected calcium (CCA) Magnesium (MAG) Glucose (GLUC) Quantitative Glucose 6-Phosphate Dehydrogenase (G6PD) (Screening only) Urea Creatinine (CREAT) Estimated glomerular filtration rate (eGFR) – CKD Epi calculation Albumin (ALB) Globulin Total protein Total protein Total bilirubin (BILI) Direct (conjugated) bilirubin (BILDIR) Alkaline phosphatase (ALP) Alanine aminotransferase (AST) Gamma-glutamyl transferase (GGT) Lactate dehydrogenase (LDH) Phosphate (PHOS) C-Reactive Protein (CRP) (not required at Screening) Cholesterol (Chol) (Screening only) Triglycerides (Trig) (Screening only) Ligh density lipoprotein (LDL) (Screening only) Low density lipoprotein (LDL) (Screening only) | Sodium (NA) |
|---|---|
| Bicarbonate (BICARB) Calcium (CA) Corrected calcium (CCA) Magnesium (MAG) Glucose (GLUC) Quantitative Glucose 6-Phosphate Dehydrogenase (G6PD) (Screening only) Urea Creatinine (CREAT) Estimated glomerular filtration rate (eGFR) – CKD Epi calculation Albumin (ALB) Globulin Total protein Total protein Total bilirubin (BILI) Direct (conjugated) bilirubin (BILDIR) Alkaline phosphatase (ALP) Alanine aminotransferase (ALT) Aspartate aminotransferase (AST) Gamma-glutamyl transferase (GGT) Lactate dehydrogenase (LDH) Phosphate (PHOS) C-Reactive Protein (CRP) (not required at Screening) Cholesterol (Chol) (Screening only) Triglycerides (Trig) (Screening only) High density lipoprotein (HDL) (Screening only) | Potassium (K) |
| Calcium (CA) Corrected calcium (CCA) Magnesium (MAG) Glucose (GLUC) Quantitative Glucose 6-Phosphate Dehydrogenase (G6PD) (Screening only) Urea Creatinine (CREAT) Estimated glomerular filtration rate (eGFR) – CKD Epi calculation Albumin (ALB) Globulin Total protein Total protein Total bilirubin (BILI) Direct (conjugated) bilirubin (BILDIR) Alkaline phosphatase (ALP) Alanine aminotransferase (ALT) Aspartate aminotransferase (AST) Gamma-glutamyl transferase (GGT) Lactate dehydrogenase (LDH) Phosphate (PHOS) C-Reactive Protein (CRP) (not required at Screening) Cholesterol (Chol) (Screening only) Triglycerides (Trig) (Screening only) High density lipoprotein (HDL) (Screening only) | Chloride (CL) |
| Corrected calcium (CCA) Magnesium (MAG) Glucose (GLUC) Quantitative Glucose 6-Phosphate Dehydrogenase (G6PD) (Screening only) Urea Creatinine (CREAT) Estimated glomerular filtration rate (eGFR) – CKD Epi calculation Albumin (ALB) Globulin Total protein Total protein Total bilirubin (BILI) Direct (conjugated) bilirubin (BILDIR) Alkaline phosphatase (ALP) Alanine aminotransferase (ALT) Aspartate aminotransferase (AST) Gamma-glutamyl transferase (GGT) Lactate dehydrogenase (LDH) Phosphate (PHOS) C-Reactive Protein (CRP) (not required at Screening) Cholesterol (Chol) (Screening only) High density lipoprotein (HDL) (Screening only) | Bicarbonate (BICARB) |
| Magnesium (MAG) Glucose (GLUC) Quantitative Glucose 6-Phosphate Dehydrogenase (G6PD) (Screening only) Urea Creatinine (CREAT) Estimated glomerular filtration rate (eGFR) – CKD Epi calculation Albumin (ALB) Globulin Total protein Total protein Total bilirubin (BILI) Direct (conjugated) bilirubin (BILDIR) Alkaline phosphatase (ALP) Alanine aminotransferase (AST) Gamma-glutamyl transferase (GGT) Lactate dehydrogenase (LDH) Phosphate (PHOS) C-Reactive Protein (CRP) (not required at Screening) Cholesterol (Chol) (Screening only) Triglycerides (Trig) (Screening only) High density lipoprotein (HDL) (Screening only) | Calcium (CA) |
| Glucose (GLUC) Quantitative Glucose 6-Phosphate Dehydrogenase (G6PD) (Screening only) Urea Creatinine (CREAT) Estimated glomerular filtration rate (eGFR) – CKD Epi calculation Albumin (ALB) Globulin Total protein Total bilirubin (BILI) Direct (conjugated) bilirubin (BILDIR) Alkaline phosphatase (ALP) Alanine aminotransferase (ALT) Aspartate aminotransferase (AST) Gamma-glutamyl transferase (GGT) Lactate dehydrogenase (LDH) Phosphate (PHOS) C-Reactive Protein (CRP) (not required at Screening) Cholesterol (Chol) (Screening only) Triglycerides (Trig) (Screening only) High density lipoprotein (HDL) (Screening only) | Corrected calcium (CCA) |
| Quantitative Glucose 6-Phosphate Dehydrogenase (G6PD) (Screening only) Urea Creatinine (CREAT) Estimated glomerular filtration rate (eGFR) – CKD Epi calculation Albumin (ALB) Globulin Total protein Total bilirubin (BILI) Direct (conjugated) bilirubin (BILDIR) Alkaline phosphatase (ALP) Alanine aminotransferase (ALT) Aspartate aminotransferase (AST) Gamma-glutamyl transferase (GGT) Lactate dehydrogenase (LDH) Phosphate (PHOS) C-Reactive Protein (CRP) (not required at Screening) Cholesterol (Chol) (Screening only) Triglycerides (Trig) (Screening only) High density lipoprotein (HDL) (Screening only) | Magnesium (MAG) |
| Urea Creatinine (CREAT) Estimated glomerular filtration rate (eGFR) – CKD Epi calculation Albumin (ALB) Globulin Total protein Total bilirubin (BILI) Direct (conjugated) bilirubin (BILDIR) Alkaline phosphatase (ALP) Alanine aminotransferase (ALT) Aspartate aminotransferase (AST) Gamma-glutamyl transferase (GGT) Lactate dehydrogenase (LDH) Phosphate (PHOS) C-Reactive Protein (CRP) (not required at Screening) Cholesterol (Chol) (Screening only) Triglycerides (Trig) (Screening only) High density lipoprotein (HDL) (Screening only) | Glucose (GLUC) |
| Creatinine (CREAT) Estimated glomerular filtration rate (eGFR) – CKD Epi calculation Albumin (ALB) Globulin Total protein Total bilirubin (BILI) Direct (conjugated) bilirubin (BILDIR) Alkaline phosphatase (ALP) Alanine aminotransferase (ALT) Aspartate aminotransferase (AST) Gamma-glutamyl transferase (GGT) Lactate dehydrogenase (LDH) Phosphate (PHOS) C-Reactive Protein (CRP) (not required at Screening) Cholesterol (Chol) (Screening only) Triglycerides (Trig) (Screening only) High density lipoprotein (HDL) (Screening only) | Quantitative Glucose 6-Phosphate Dehydrogenase (G6PD) ( <i>Screening only</i> ) |
| Estimated glomerular filtration rate (eGFR) – CKD Epi calculation Albumin (ALB) Globulin Total protein Total bilirubin (BILI) Direct (conjugated) bilirubin (BILDIR) Alkaline phosphatase (ALP) Alanine aminotransferase (ALT) Aspartate aminotransferase (AST) Gamma-glutamyl transferase (GGT) Lactate dehydrogenase (LDH) Phosphate (PHOS) C-Reactive Protein (CRP) (not required at Screening) Cholesterol (Chol) (Screening only) Triglycerides (Trig) (Screening only) High density lipoprotein (HDL) (Screening only) | Urea |
| Albumin (ALB) Globulin Total protein Total bilirubin (BILI) Direct (conjugated) bilirubin (BILDIR) Alkaline phosphatase (ALP) Alanine aminotransferase (ALT) Aspartate aminotransferase (AST) Gamma-glutamyl transferase (GGT) Lactate dehydrogenase (LDH) Phosphate (PHOS) C-Reactive Protein (CRP) (not required at Screening) Cholesterol (Chol) (Screening only) Triglycerides (Trig) (Screening only) High density lipoprotein (HDL) (Screening only) | |
| Globulin Total protein Total bilirubin (BILI) Direct (conjugated) bilirubin (BILDIR) Alkaline phosphatase (ALP) Alanine aminotransferase (ALT) Aspartate aminotransferase (AST) Gamma-glutamyl transferase (GGT) Lactate dehydrogenase (LDH) Phosphate (PHOS) C-Reactive Protein (CRP) (not required at Screening) Cholesterol (Chol) (Screening only) Triglycerides (Trig) (Screening only) High density lipoprotein (HDL) (Screening only) | Estimated glomerular filtration rate (eGFR) – CKD Epi calculation |
| Total protein Total bilirubin (BILI) Direct (conjugated) bilirubin (BILDIR) Alkaline phosphatase (ALP) Alanine aminotransferase (ALT) Aspartate aminotransferase (AST) Gamma-glutamyl transferase (GGT) Lactate dehydrogenase (LDH) Phosphate (PHOS) C-Reactive Protein (CRP) (not required at Screening) Cholesterol (Chol) (Screening only) Triglycerides (Trig) (Screening only) High density lipoprotein (HDL) (Screening only) | |
| Total bilirubin (BILI) Direct (conjugated) bilirubin (BILDIR) Alkaline phosphatase (ALP) Alanine aminotransferase (ALT) Aspartate aminotransferase (AST) Gamma-glutamyl transferase (GGT) Lactate dehydrogenase (LDH) Phosphate (PHOS) C-Reactive Protein (CRP) (not required at Screening) Cholesterol (Chol) (Screening only) Triglycerides (Trig) (Screening only) High density lipoprotein (HDL) (Screening only) | |
| Direct (conjugated) bilirubin (BILDIR) Alkaline phosphatase (ALP) Alanine aminotransferase (ALT) Aspartate aminotransferase (AST) Gamma-glutamyl transferase (GGT) Lactate dehydrogenase (LDH) Phosphate (PHOS) C-Reactive Protein (CRP) (not required at Screening) Cholesterol (Chol) (Screening only) Triglycerides (Trig) (Screening only) High density lipoprotein (HDL) (Screening only) | |
| Alkaline phosphatase (ALP) Alanine aminotransferase (ALT) Aspartate aminotransferase (AST) Gamma-glutamyl transferase (GGT) Lactate dehydrogenase (LDH) Phosphate (PHOS) C-Reactive Protein (CRP) (not required at Screening) Cholesterol (Chol) (Screening only) Triglycerides (Trig) (Screening only) High density lipoprotein (HDL) (Screening only) | $\lambda = I$ |
| Alanine aminotransferase (ALT) Aspartate aminotransferase (AST) Gamma-glutamyl transferase (GGT) Lactate dehydrogenase (LDH) Phosphate (PHOS) C-Reactive Protein (CRP) (not required at Screening) Cholesterol (Chol) (Screening only) Triglycerides (Trig) (Screening only) High density lipoprotein (HDL) (Screening only) | |
| Aspartate aminotransferase (AST) Gamma-glutamyl transferase (GGT) Lactate dehydrogenase (LDH) Phosphate (PHOS) C-Reactive Protein (CRP) (not required at Screening) Cholesterol (Chol) (Screening only) Triglycerides (Trig) (Screening only) High density lipoprotein (HDL) (Screening only) | |
| Gamma-glutamyl transferase (GGT) Lactate dehydrogenase (LDH) Phosphate (PHOS) C-Reactive Protein (CRP) (not required at Screening) Cholesterol (Chol) (Screening only) Triglycerides (Trig) (Screening only) High density lipoprotein (HDL) (Screening only) | |
| Lactate dehydrogenase (LDH) Phosphate (PHOS) C-Reactive Protein (CRP) (not required at Screening) Cholesterol (Chol) (Screening only) Triglycerides (Trig) (Screening only) High density lipoprotein (HDL) (Screening only) | |
| Phosphate (PHOS) C-Reactive Protein (CRP) (not required at Screening) Cholesterol (Chol) (Screening only) Triglycerides (Trig) (Screening only) High density lipoprotein (HDL) (Screening only) | Gamma-glutamyl transferase (GGT) |
| C-Reactive Protein (CRP) (not required at Screening) Cholesterol (Chol) (Screening only) Triglycerides (Trig) (Screening only) High density lipoprotein (HDL) (Screening only) | |
| Cholesterol (Chol) ( <i>Screening only</i> ) Triglycerides (Trig) ( <i>Screening only</i> ) High density lipoprotein (HDL) ( <i>Screening only</i> ) | |
| Triglycerides (Trig) ( <i>Screening only</i> ) High density lipoprotein (HDL) ( <i>Screening only</i> ) | |
| High density lipoprotein (HDL) (Screening only) | |
| Low density lipoprotein (LDL) ( <i>Screening only</i> ) | |
| | Low density lipoprotein (LDL) ( <b>Screening only</b> ) |

### Pregnancy Test and FSH

β-Human Chorionic Gonadotropin (β-HCG) (women of child bearing potential only)

BM S01-A, v3.0

Statistical Analysis Plan Effective: 17/SEP/2020 CONFIDENTIAL


Follicular Stimulating Hormone (FSH) (post-menopausal women only)

### **Urinalysis**

| Glucose (GLUC) |
|------------------------------------------------------------------------------|
| Bilirubin (BILI) |
| Ketone (KETONES) |
| Specific gravity (SPGRAV) |
| Blood |
| рН |
| Protein (PROT) |
| Urobilinogen (UROBIL) |
| Nitrite |
| Leukocytes (WBC) |
| Microscopy, culture and sensitivity (formal laboratory analysis if required) |

### Coagulation

| Prothrombin Time (PT) |
|----------------------------------------------|
| Activated Partial Thromboplastin Time (APTT) |
| International Normalised Ratio (INR) |

### Viral Screen

| HIV 1/2 (anti-HIV1 and anti-HIV2 Ab) |
|--------------------------------------------------------------|
| Hepatitis B (HBsAg, anti-HBc [IgG + IgM if IgG is positive]) |
| Hepatitis C (anti-HCV) |

### Biostatistical methods

### Listings

All laboratory parameters and change from treatment baseline values will be presented in data listings. Values outside the laboratory reference range will be listed with flags if considered low or high for values outside the reference ranges (where applicable) and if values considered to be clinically significant by the investigator.

Pregnancy test data will be listed only, for all women. FSH data will be listed only, for all post-menopausal women.

Coagulation data as well as qualitative and quantitative urinalysis data will also be listed only.

#### Tables

Haematology, biochemistry and continuous dipstick urinalysis laboratory data will be summarised for each scheduled visit, including observed values, absolute change from treatment baseline.

Categorical dipstick urinalysis results will be summarised for each scheduled visit using frequency tabulations.

BM S01-A, v3.0

Statistical Analysis Plan


Effective: 17/SEP/2020 


Numbers of participants with treatment-emergent abnormalities will also be shown.

### 11.3.4 Vital Signs

#### **Parameters**

- Systolic Blood Pressure (SBP) (mmHg)
- Diastolic Blood Pressure (DBP) (mmHg)
- Heart Rate (beats/minute)
- Body Temperature (°C)
- Respiratory rate (beats/min)

#### Biostatistical methods

All vital signs data will be listed for all participants. Any values outside of the protocol defined normal ranges will be flagged, with clinical significance status presented for out-of-range results.

Table 1: Vital Signs Normal Ranges

| Parameter | Range |
|--------------------------|-------------------|
| Systolic blood pressure | 90-140 mmHg |
| Diastolic blood pressure | 50-90 mmHg |
| Heart rate | 50-100 bpm |
| Temperature | 35.0-37.5°C |
| Respiratory rate | 10-25 breaths/min |

Vital sign parameters will be summarised by presenting summary statistics for observed values and change from treatment baseline values for each scheduled visit.

### 11.3.5 Body Measurements

#### Definition of variables

- Height (Screening Only)
- Weight
- Body mass index (BMI)

#### Biostatistical methods

Body measurement data will be listed for all participants and visits, including height, weight and Body Mass Index (BMI) which is auto-calculated within the CRF.

Observed values, as well as changes from treatment baseline, will be summarised descriptively for weight and BMI by visit.

### 11.3.6. Physical Examination

#### **Parameters**

- Weight
- HEENT (Head, Eyes, Ears, Nose, Throat)
- Height (screening only)
- Chest / Lungs
- Abdomen

- Skin
- Neurological / Reflexes
- Heart / circulation
- Neck

BM S01-A, v3.0

Statistical Analysis Plan


#### Biostatistical methods

Physical examination findings will be listed for all participants and visits.

#### 11.3.7. 12-lead ECG

#### **Parameters**

- PR interval (msec)
- QRS interval (msec)
- QTcF interval (msec)
- Overall ECG assessment (Normal, Abnormal)
- ECG abnormality (specify as appropriate)
- Clinical Significance

### Biostatistical methods

ECG parameters will be listed for all participants and visits. Triplicate ECGs will be presented in listings for individual readings as well as the mean for each triplicate. The triplicate means will be used for the summary table. Any values outside of the protocol defined normal ranges (Table XX) will be flagged.

Table 2: ECG Normal Ranges

| Parameter | Range |
|-------------|--------------------|
| PR interval | ≤210 msec |
| QRS | 50-120 msec |
| QTcF | Males: ≤450 msec |
| | Females: ≤470 msec |

Observed values, as well as changes from treatment baseline, will be summarised descriptively for all ECG parameters by visit. An addition table will present the frequencies of participants who fulfill the following prolongation (change from baseline) criteria, considering all scheduled and non-scheduled visit data:

- QTcF prolongation >30
- QTcF prolongation >60
- QTcF >450 msec for males
- QTcF >450 msec for females
- QTcF >470 msec for females

### 11.3.8. Malaria Clinical Score

Malaria clinical score data will be listed for all participants, including the individual scores for each of the 14 signs/symptoms as well as the total score.

The number (and percentage) of participants scoring each symptom (0=absent; 1=mild; 2=moderate; 3=severe) will be tabulated per dose group and per protocol defined timepoint.

The highest score as well as the time(s) to the highest score observed will be tabulated.

### 11.3.9. Presentation of Safety Results

The table summary and listings of AEs and lab parameters will be presented for the CSR, and are provided in Appendix, Table B.


BM S01-A, v3.0

Statistical Analysis Plan 


#### 12. EXPLORATORY PARAMETERS

Analysis Set: PD Analysis Set

Endpoint: Incidence and level of resistance to MMV367 in parasites determined using *in vitro* methods.

Parasites will be genotyped and in vitro drug sensitivity testing will be performed.

Endpoint: Effect of MMV367 on parasite viability in ex vivo cultures.

Ex vivo growth is a measure of parasite viability. An estimate of the number of viable parasites following MMV367 treatment will be quantified using a limiting dilution assay by counting the number of wells with parasite growth using the following formula [8]:

$$Viable\ parasites = X^{n-1},$$

Where n is the number of wells with parasite growth and X is the dilution factor used in the assay. If no wells exhibit parasite growth (i.e. n=0) the number of viable parasites is estimated to be zero. Short term ex vivo cultures will be established from blood samples collected pre-MMV367 administration (Day 8), then at several time-points post-MMV367 administration. An estimate of the number of initial parasites will be established using the pre-MMV367 administration samples, which will be used to calculate a normalization factor for post-MMV367 administration samples. Limiting dilution assays will be run for participant samples in triplicate, with the estimate of the number of viable parasites described for each sample as a mean (SD) on the log-scale. Estimates of both the raw number of viable parasites and the normalized number of viable parasites will be presented. Estimates of viable parasites may also be summarized by MMV367 dose per study time-point, with dose comparisons assessed using ANOVA, Kruskal Wallis tests or equivalent, as appropriate. The results of parasite ex vivo growth analyses will be supportive to malaria 18S qPCR data in determining the kinetics of parasite clearance following MMV367 dosing (secondary endpoint).

### 13. CHANGES TO THE PLANNED ANALYSIS

There is no change to the planned analysis by the time this SAP was written.

#### 14. INTERIM AND FINAL ANALYSIS

This study has no formal interim analyses other than review of safety, tolerability, parasitaemia and PK parameters by the SDRT between cohorts.

### 15. SOFTWARE

SAS® Version 9.4 or higher (SAS Institute, Cary, North Carolina, USA) for Safety, demographic and baseline characteristics, participant disposition, protocol deviations, prior medications and treatment exposure analyses

All PK/PD analyses will be performed in R 4.1.3 and IQRtool package 1.10.0 [IQRtools]. NLME modelling will be performed with Monolix 2019R1 [MLX19] using Stochastic Approximation Expectation Maximization (SAEM) for parameter estimation. For PD modelling where typically the variance of random effects cannot be estimated

BM S01-A, v3.0

Statistical Analysis Plan


from the data, the IQRtools SysFit approach [KAS19] will be used to estimate typical and individual PD parameters.

Data manipulation and data analyses for all pharmacodynamic data will be performed using R (highest version available).

### 16. REFERENCES

- 1) Wang CYT, Ballard EL, Pava Z Marquart L, Gaydon J, Murphy SC, Whiley D, O'Rourke P, McCarthy JS (2021) Analytical validation of a real-time hydrolysis probe PCR assay for quantifying Plasmodium falciparum parasites in experimentally infected human adults, *Malaria Journal*, 20(181).
- 2) Marquart L, Baker M, O'Rourke P, McCarthy JS (2015) Evaluating the pharmacodynamic effect of antimalarial drugs in clinical trials by quantitative PCR, *Antimicrobrial Agents and Chemotherapy*, 59, 4249–59.
- 3) IQRtools https://www.intiquan.com/iqr-tools/
- 4) **KAS19** Kaschek D, Mader W, Fehling-Kaschek M, Rosenblatt M, Timmer J. Dynamic Modeling, Parameter Estimation, and Uncertainty Analysis in R. J. Stat. Soft. 2019 Apr 30;88(10):1-32.
- 5) **RAU09** Raue A, Kreutz C, Maiwald T, Bachmann J, Schilling M, Klingmüller U, Timmer J. Structural and practical identifiability analysis of partially observed dynamical models by exploiting the profile likelihood. Bioinformatics. 2009 Jun 8;25(15):1923-9.
- 6) MMV MMV367 protocol FINAL v2.0 14Apr23 Clean signed.
- 7) eCOS UniqueCRFs UniquePages MMV 367 22 01 2023-04-17
- 8) Sanz LM, Crespo B, De-Cózar C, Ding XC, Llergo JL, Burrows JN, García-Bustos JF, Gamo FJ. P. falciparum in vitro killing rates allow to discriminate between different antimalarial mode-of-action. PLoS One. 2012;7(2):e30949. doi: 10.1371/journal.pone.0030949. Epub 2012 Feb 23. PMID: 22383983; PMCID: PMC3285618.

### 17. APPENDIX

Table A. PD and PK Planned Tables, Listings and Figures

| Title | Analysis Set |
|---------------------------------------------|--------------|
| PD Listings | |
| Pharmacodynamic –Parasitemia | PD |
| Pharmacodynamic –Parasite Life Cycle Stages | PD |
| PK Listings | |
| Pharmacokinetic Concentrations | PK |
| Pharmacokinetic Parameters | PK |
| PD Tables | |
| Summary of Malaria Parasitaemia (18S qPCR) | PD |

BM S01-A, v3.0

Statistical Analysis Plan CONFIDENTIAL

| Summary of Malaria Parasite Lifecycle Stage Data (pfs25. pfMGET and SBP-1 qRT-PCR) | PD |
|---|---|
| PK Tables | |
| Summary of Pharmacokinetic Concentration | PK |
| Summary of Pharmacokinetic Parameters | PK |
| PD Figures | |
| Individual qPCR 18s-time Profiles | PD |
| Individual RT-PCR pfs25-time Profiles | PD |
| Individual RT-PCR pfMGET-time Profiles | PD |
| Individual RT-PCR SBP-1-time Profiles | PD |
| PK Figures | |
| Arithmetic Mean (+SD) Pharmacokinetic Concentration-time Profiles by Dose Group | PK |
| Individual Pharmacokinetic Concentration-time Profiles | PK |

Table B. Baseline Characteristics and Safety Analysis Tables and Listings

| Title | Analysis Set |
|--------------------------------------------------------------|--------------|
| Listings | |
| Participant Disposition | FAS |
| Dose Group Assignment | FAS |
| Protocol Deviations | FAS |
| Analysis Population Assignment | FAS |
| Demographics | FAS |
| Medical History | FAS |
| Pregnancy Test | FAS |
| Follicle Stimulating Hormone (FSH) | FAS |
| Viral Screen | FAS |
| Urine Drug Screening | FAS |
| Alcohol Breath Test | FAS |
| Positive SARS-CoV-2 | FAS |
| Prior Medications | |
| Concomitant Medications | FAS |
| Inoculum Administration | FAS |
| IMP Administration | FAS |
| Rescue Medication Administration | FAS |
| Inoculum-Emergent Adverse Events | FAS |
| Treatment-Emergent Adverse Events | IMP |
| Inoculum related Inoculum-Emergent Adverse Events | FAS |
| IMP related Treatment-Emergent Adverse Events | IMP |
| Inoculum Emergent Serious Adverse Events | FAS |
| Treatment Emergent Serious Adverse Events | IMP |
| Inoculum-Emergent Adverse Events Leading to Discontinuation | FAS |
| Treatment-Emergent Adverse Events Leading to Discontinuation | IMP |
| Inoculum-Emergent Adverse Events of Special Interest | FAS |
| Treatment-Emergent Adverse Events of Special Interest | IMP |

BM S01-A, v3.0

CONFIDENTIAL Statistical Analysis Plan

| Deaths | TAC |
|---|---|
| Deaths | FAS |
| Individual Haematology Results | FAS |
| Individual Biochemistry Results | FAS |
| Coagulation Screening | FAS |
| Individual Urinalysis Results (dipstick) | FAS |
| Individual Urine Microscopy Results | FAS |
| Individual Vital Signs Results | FAS |
| Individual ECG Parameters Results | FAS |
| Physical Examination | FAS |
| Malaria Clinical Score Results | FAS |
| Tables | |
| Analysis Populations | FAS |
| Participant Disposition | FAS |
| Demographics and Baseline Characteristics | FAS |
| Summary of Prior Medications | FAS |
| Protocol Deviations | FAS |
| Overall Summary of Inoculum Emergent Adverse Events | FAS |
| Overall Summary of Treatment Emergent Adverse Events | IMP |
| Summary of Inoculum Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (All Causalities) | FAS |
| Summary of Treatment Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (All Causalities) | IMP |
| Summary of Inoculum Emergent Adverse Events by Maximum Severity (All Causalities) | FAS |
| Summary of Treatment Emergent Adverse Events by Maximum Severity (All Causalities) | IMP |
| Summary of Inoculum related Treatment Emergent Adverse Events by MedDRA System Organ Class, Preferred Term | FAS |
| Summary of IMP Related Treatment Emergent Adverse Events by MedDRA System Organ Class, Preferred Term | IMP |
| Summary of Inoculum Related IEAEs by System Organ Class, Preferred Term and Maximum Severity | FAS |
| Summary of IMP Related TEAEs by System Organ Class, Preferred Term and Maximum Severity | IMP |
| Inoculum Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term (All Causalities) | FAS |
| Treatment Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term (All Causalities) | IMP |
| Overall Summary of Inoculum Emergent Adverse Events of Special Interest (AESI) | FAS |
| Overall Summary of Treatment Emergent Adverse Events of Special Interest (AESI) | IMP |
| Inoculum Emergent Adverse Events of Special Interest (AESI) by MedDRA System Organ Class and Preferred Term (All Causalities) | FAS |
| Treatment Emergent Adverse Events of Special Interest (AESI) by MedDRA System Organ Class and Preferred Term (All Causalities) | IMP |
| Inoculum Emergent Adverse Events Leading to Study Discontinuation by MedDRA System Organ Class and Preferred Term (All Causalities) | FAS |
| Treatment Emergent Adverse Events Leading to Study Discontinuation by MedDRA System Organ Class and Preferred Term (All Causalities) | IMP<br>FAS |
| Summary of Concomitant Medications (FAS) | |
| Summary of Concomitant Medications (IMP) | IMP |
| Haematology (Summary and Change from IMP Baseline) | FAS |
| Haematology (Categorical) | FAS |
| Biochemistry (Summary and Change from IMP Baseline) | FAS |
| Biochemistry (Categorical) | FAS |
| Urinalysis (Continuous) Results and Change from Baseline | FAS |
| Urinalysis (Categorical) Results | FAS |

| Vital Signs Results and Change from IMP Baseline | FAS |
|---|---|
| Abnormal Vital Signs Results | FAS |
| ECG Results and Change from IMP Baseline | FAS |
| ECG QTc Categorical Analyses | FAS |
| ECG Clinical Assessment | FAS |
| Malaria Clinical Score Summary by Question | FAS |
| Summary Peak Total Malaria Clinical Score and Time to Peak Total Malaria Clinical Score | FAS |

BM S01-A, v3.0

CONFIDENTIAL Statistical Analysis Plan